CLINICAL TRIAL: NCT03201419
Title: A Randomised, Double-blind, Placebo-controlled, Response-adaptive Dose-finding Trial Investigating the Efficacy, Safety and Tolerability of Oral Doses of FE 201836, With Desmopressin Orally Disintegrating Tablet as a Benchmark, During 12 Weeks of Treatment for Nocturia Due to Nocturnal Polyuria in Adults
Brief Title: A Trial to Investigate Efficacy, Safety and Tolerability of FE 201836 for Nocturia Due to Nocturnal Polyuria in Adults
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Ferring Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 000233; 2016-003851-31 (EudraCT Number)
Record Dates: First submitted 2017-06-26; First posted 2017-06-28 (Actual); Results first posted 2020-12-23 (Actual); Last update posted 2022-03-02 (Actual); Status verified 2020-10

CONDITIONS: Nocturia
MeSH Terms: conditions — Nocturia | interventions — Deamino Arginine Vasopressin

STUDY DESIGN:
Intervention Model Description: The trial consisted of a 2 week period of screening/lifestyle changes during which no treatment was given, a 2 week enrichment period (including a 1 week single blind active run-in period [FE 201836 500 µg] and a 1 week washout period) followed by a 12 week randomized treatment period for each subject. Prior to the first interim analysis, the first 129 subjects were randomized to daily treatment with FE 201836 500 µg, placebo, or desmopressin (25 µg for females and 50 µg for males) in a 2:2:1 ratio. After the first interim analysis, subjects were randomized to daily treatment with FE 201836 (50 µg, 100 µg, 150 µg, 250 µg, 350 µg, or 500 µg), placebo, or desmopressin (25 µg for females and 50 µg for males) using response adaptive allocation probabilities.
Who Masked: Participant, Investigator
Masking Description: Each subject will receive 2 medications (an oral solution and an orally disintegrating tablet (ODT) formulation) throughout the trial, in order to keep the treatment blinded.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (9):
- FE 201836 500 μg (Randomized Treatment Period) (Experimental): FE 201836 500 μg oral solution and placebo orally disintegrating tablet (ODT), administered once daily
  Interventions: Drug: FE 201836; Drug: Placebo ODT
- FE 201836 350 μg (Randomized Treatment Period) (Experimental): FE 201836 350 μg oral solution and placebo ODT, administered once daily
  Interventions: Drug: FE 201836; Drug: Placebo ODT
- FE 201836 250 μg (Randomized Treatment Period) (Experimental): FE 201836 250 μg oral solution and placebo ODT, administered once daily
  Interventions: Drug: FE 201836; Drug: Placebo ODT
- FE 201836 150 μg (Randomized Treatment Period) (Experimental): FE 201836 150 μg oral solution and placebo ODT, administered once daily
  Interventions: Drug: FE 201836; Drug: Placebo ODT
- FE 201836 100 μg (Randomized Treatment Period) (Experimental): FE 201836 100 μg oral solution and placebo ODT, administered once daily
  Interventions: Drug: FE 201836; Drug: Placebo ODT
- FE 201836 50 μg (Randomized Treatment Period) (Experimental): FE 201836 50 μg oral solution and placebo ODT, administered once daily
  Interventions: Drug: FE 201836; Drug: Placebo ODT
- Placebo (Randomized Treatment Period) (Experimental): Placebo oral solution and placebo ODT, administered once daily
  Interventions: Drug: Placebo oral solution; Drug: Placebo ODT
- Desmopressin 25 μg (Randomized Treatment Period) (Experimental): Desmopressin 25 μg ODT and placebo oral solution, administered once daily (female subjects)
  Interventions: Drug: Desmopressin; Drug: Placebo oral solution
- Desmopressin 50 μg (Randomized Treatment Period) (Experimental): Desmopressin 50 μg ODT and placebo oral solution, administered once daily (male subjects)
  Interventions: Drug: Desmopressin; Drug: Placebo oral solution

INTERVENTIONS:
Drug: FE 201836 — Oral solution for daily intake
  Other Names: Velmupressin
  Arms: FE 201836 100 μg (Randomized Treatment Period); FE 201836 150 μg (Randomized Treatment Period); FE 201836 250 μg (Randomized Treatment Period); FE 201836 350 μg (Randomized Treatment Period); FE 201836 50 μg (Randomized Treatment Period); FE 201836 500 μg (Randomized Treatment Period)
Drug: Desmopressin — Desmopressin Orally Disintegrating Tablet (ODT)
  Other Names: NOCDURNA
  Arms: Desmopressin 25 μg (Randomized Treatment Period); Desmopressin 50 μg (Randomized Treatment Period)
Drug: Placebo oral solution — Manufactured to mimic experimental drug
  Arms: Desmopressin 25 μg (Randomized Treatment Period); Desmopressin 50 μg (Randomized Treatment Period); Placebo (Randomized Treatment Period)
Drug: Placebo ODT — Manufactured to mimic experimental drug
  Arms: FE 201836 100 μg (Randomized Treatment Period); FE 201836 150 μg (Randomized Treatment Period); FE 201836 250 μg (Randomized Treatment Period); FE 201836 350 μg (Randomized Treatment Period); FE 201836 50 μg (Randomized Treatment Period); FE 201836 500 μg (Randomized Treatment Period); Placebo (Randomized Treatment Period)

SUMMARY:
The purpose of this trial was to investigate the efficacy, safety and tolerability of different oral doses of FE 201836, with desmopressin as a benchmark, during 12 weeks of treatment for nocturia due to nocturnal polyuria in adults

ELIGIBILITY:
Inclusion Criteria:

* Adults ≥18 years of age (at the time of written consent)
* Medical history of, or subject reported nocturia symptoms during the 6 months prior to Visit 1
* ≥2 nocturnal voids (an average over 3 days) as documented in the 3-day e-Diary prior to Visit 2
* The largest single voided volume must be ≥200 mL (at least 1 void ≥200 mL) as documented in the 3-day e-Diary prior to Visit 2
* Nocturnal polyuria, defined as Nocturnal Polyuria index >33%, a ratio of Nocturnal Urine Volume in excess of 33% of total daily (24-hour) urine volume as documented in the 3-day e-Diary prior to Visit 2
* ≥20% decrease in the nocturnal diuresis rate (mL/min) (that was recorded at Visit 2) as documented in the 3-day e-Diary prior to Visit 3

Exclusion Criteria:

* Current diagnosis of Obstructive Sleep Apnoea (OSA)
* Restless Legs Syndrome (RLS)
* Bladder Outlet Obstruction (BOO) or urine flow <5 mL/s, as confirmed by uroflowmetry upon suspicion during screening prior to Visit 2
* Urinary incontinence defined as an average of >1 episode/day in the 3-day e-Diary prior to Visit 2 (occasional urge incontinence during daytime or at night on the way to void is not necessarily exclusionary)
* Any pelvic or lower urinary tract surgery and/or radio therapy or previous pelvic irradiation within the past 6 months prior to Visit 1. Including e.g., transurethral resection for Bladder Outlet Obstruction or Benign Prostatic Hyperplasia, hysterectomy or female incontinence procedures
* Genito-urinary tract pathology that can in the investigator's opinion be responsible for urgency or urinary incontinence e.g., symptomatic or recurrent urinary tract infections, interstitial cystitis, bladder-related pain, chronic pelvic pain syndrome, or stone in the bladder or urethra causing symptoms
* A history of cancer with the last date of disease activity/presence of malignancy within the last 12 months prior to Visit 1, except for adequately treated basal cell carcinoma of the skin
* History of any neurological disease affecting bladder function or muscle strength (e.g., Multiple Sclerosis, Parkinson's, spinal cord injury, spina bifida)
* Habitual (fluid intake >3L per day) or psychogenic polydipsia
* Uncontrolled hypertension, as judged by the investigator
* Uncontrolled diabetes mellitus, as judged by the investigator
* Central or nephrogenic diabetes insipidus
* Known history of Syndrome of Inappropriate Antidiuretic Hormone (SIADH) secretion
* History of gastric retention
* Suspicion or evidence of congestive heart failure, (New York Heart Association (NYHA) class II, III, IV)
* Hyponatraemia:

  * Serum sodium level <135 mmol/L at Visit 1(re-tested, with results available within 7 days)
  * Serum sodium level <130 mmol/L at Visit 3 (re-tested, with results available within 7 days)
* Use of any prohibited therapy listed below:

  * Current or former (within 3 months prior to screening) treatment with any other investigational medicinal product (IMP)
  * Unstable electrostimulation or behavioural bladder training program less than 3 months prior to screening (stable electrostimulation or behavioural bladder training program started at least 3 months before screening are acceptable)
  * Thiazide diuretics
  * Antiarrhythmic agents
  * V2-receptor antagonists/agonists (e.g., vaptans/desmopressin, vasopressin)
  * Loperamide
  * Botulinum toxin (cosmetic non-urological use is acceptable)
  * Valproate

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 302 (Actual)
Dates: Start 2017-07-27 (Actual); Primary Completion 2019-10-31 (Actual); Study Completion 2019-10-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Compliance, Study Director — Ferring Pharmaceuticals
Locations (72):
- United States (43):
  - Achieve Clinical Research, LLC, Birmingham, Alabama
  - Coastal Clinical Research, an AMR company, Mobile, Alabama
  - Clinical Trials Research, Lincoln, California
  - Tri Valley Urology Medical Group, Murrieta, California
  - San Diego Clinical Trials, San Diego, California
  - Advanced Rx Clinical Research Group, Inc., Westminster, California
  - Downtown Women's Health Care, Denver, Colorado
  - Genitourinary Surgical Consultants, P.C., Denver, Colorado
  - South Florida Medical Research, Aventura, Florida
  - Women's Medical Research Group, LLC, Clearwater, Florida
  - Tampa Bay Medical Research, Inc., Clearwater, Florida
  - Clinical Research of South Florida, Coral Gables, Florida
  - Avail Clinical Research, LLC, DeLand, Florida
  - Finlay Medical Research Corp, Greenacres City, Florida
  - Pharmax Research Clinic, Miami, Florida
  - Doctors Research Institute Corporation, Miami, Florida
  - Sanitas Research, Miami, Florida
  - Bayside Clinical Research LLC, New Port Richey, Florida
  - Pines Care Research Center, Inc, Pembroke Pines, Florida
  - Clinical Research Center of Florida, Pompano Beach, Florida
  - Meridien Research, Inc., St. Petersburg, Florida
  - American Health Network of Indiana, LLC, Avon, Indiana
  - American Health Network of Indiana, LLC, Greenfield, Indiana
  - Bay State Clinical Trials, Inc., Watertown, Massachusetts
  - Beyer Research, Kalamazoo, Michigan
  - Remedica LLC, Rochester, Michigan
  - Quality Clinical Research Center, Inc., Omaha, Nebraska
  - Clinical Research Consortium, an AMR company, Las Vegas, Nevada
  - Mid Hudson Medical Research, PLLC, New Windsor, New York
  - Premier Medical Group of the Hudson Valley, PC, Poughkeepsie, New York
  - American Health Research, Inc., Charlotte, North Carolina
  - Medication Management, LLC, Greensboro, North Carolina
  - Peters Medical Research, High Point, North Carolina
  - PMG Research of Raleigh, LLC, Raleigh, North Carolina
  - PMG Research of Wilmington, LLC, Wilmington, North Carolina
  - HWC Women's Research Center, Englewood, Ohio
  - NECCR Primacare Research, LLC, Providence, Rhode Island
  - Coastal Carolina Research Center, Inc, Mt. Pleasant, South Carolina
  - PMG Research of Charleston, LLC, Mt. Pleasant, South Carolina
  - MCA Research - Partner, Houston, Texas
  - Ericksen Research & Development, LLC, Clinton, Utah
  - Advanced Research Institute, Ogden, Utah
  - Clinical Research Associates of Tidewater, an AMR company, Norfolk, Virginia
- Belgium (5):
  - ULB Hopital Erasme, Brussels
  - UZ Antwerpen, Edegem
  - Universitair Ziekenhuis Gent, Ghent
  - AZ Groeninge - Campus Vercruysselaan, Kortrijk
  - UZ Leuven, Leuven
- Canada (10):
  - Ultra-Med Inc., Pointe-Claire, Quebec
  - Milestone Research, London
  - SKDS Research Inc., Newmarket
  - Clinique Médicale St-Louis (Recherche) inc d/b/a/ Centre de Recherche Saint-Louis, Québec
  - DIEX Recherche Quebec Inc., Québec
  - Bluewater Health-Norman Site, Sarnia
  - CHUS - Hôpital Fleurimont, Sherbrooke
  - DIEX Recherche Sherbrooke Inc., Sherbrooke
  - Ferring Investigational Site, Toronto
  - DIEX Recherche Victoriaville Inc., Victoriaville
- Czechia (5):
  - Urologie Benešov - Afimed s.r.o., Benešov
  - Fakultni nemocnice Brno, Dept of Klinika nemoci plicnich a tuberkulozy, Brno
  - Krajska nemocnice Liberec, a.s., Liberec
  - Urocentrum Plzen, Pilsen
  - Thomayerova nemocnice, PARENT, Prague
- Germany (3):
  - Gemeinschaftspraxis fuer Urologie und Andrologie, Duisburg
  - Urologische Gemeinschaftspraxis, Emmendingen
  - Klinikum Weiden, Klinik f. Urologie, Andrologie und Kinderurologie, Weiden
- Hungary (5):
  - Jahn Ferenc Del-pesti Korhaz es Rendelointezet, Budapest
  - Synexus Magyarorszag Kft., Budapest
  - Bagoly Egeszseghaz, Kecskemét
  - SzSzB Megyei Korhazak es Egyetemi Oktatokorhaz, Josa Andras Oktatokorhaz Urologia, Nyíregyháza
  - Jasz-Nagykun-Szolnok Megyei Hetenyi Geza Korhaz-Rendelointezet, Szolnok
- Nasz Lekarz Osrodek Badan Klinicznych, Bydgoszcz, Poland

REFERENCES:
- [Background] Hudgens S, Howerter A, Polek E, Andersson FL. Psychometric validation and interpretation of the Nocturia Impact Diary in a clinical trial setting. Qual Life Res. 2022 Jun;31(6):1837-1848. doi: 10.1007/s11136-021-03060-4. Epub 2021 Dec 21. PMID 34932192

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 71 sites were authorized to recruit subjects for the trial between July 2017 and July 2019. The trial sites that screened subjects to the trial were: 5 in Belgium, 10 in Canada, 5 in Czech Republic, 2 in Germany, 5 in Hungary, 1 in Poland and 43 in the Unites States of America (USA).
Pre-assignment Details: A total of 1721 subjects were screened, wherein, 531 met the eligibility criteria and entered the enrichment period. Of these, 302 subjects met the eligibility criteria at Visit (V) 4 (randomization), and were randomized to treatment with FE 201836 (different doses), placebo, or desmopressin. A total of 278 subjects completed the trial.
Groups:
- FE 201836 500 µg (Randomized Treatment Period): FE 201836 500 µg oral solution and placebo orally disintegrating tablet (ODT), administered once daily
- FE 201836 350 µg (Randomized Treatment Period): FE 201836 350 µg oral solution and placebo ODT, administered once daily
- FE 201836 250 µg (Randomized Treatment Period): FE 201836 250 µg oral solution and placebo ODT, administered once daily
- FE 201836 150 µg (Randomized Treatment Period): FE 201836 150 µg oral solution and placebo ODT, administered once daily
- FE 201836 100 µg (Randomized Treatment Period): FE 201836 100 µg oral solution and placebo ODT, administered once daily
- FE 201836 50 µg (Randomized Treatment Period): FE 201836 50 µg oral solution and placebo ODT, administered once daily
- Desmopressin 25 µg (Randomized Treatment Period): Desmopressin 25 µg ODT and placebo oral solution, administered once daily (female subjects)
- Desmopressin 50 µg (Randomized Treatment Period): Desmopressin 50 µg ODT and placebo oral solution, administered once daily (male subjects)
Period: Overall Study
Arm/Group | FE 201836 500 µg (Randomized Treatment Period) | FE 201836 350 µg (Randomized Treatment Period) | FE 201836 250 µg (Randomized Treatment Period) | FE 201836 150 µg (Randomized Treatment Period) | FE 201836 100 µg (Randomized Treatment Period) | FE 201836 50 µg (Randomized Treatment Period) | Placebo (Randomized Treatment Period) | Desmopressin 25 µg (Randomized Treatment Period) | Desmopressin 50 µg (Randomized Treatment Period)
Started | 60 | 27 | 24 | 14 | 13 | 34 | 87 | 26 | 17
Completed | 52 | 24 | 22 | 14 | 12 | 33 | 81 | 25 | 15
Not Completed | 8 | 3 | 2 | 0 | 1 | 1 | 6 | 1 | 2
Not completed — Adverse Event | 3 | 1 | 0 | 0 | 1 | 1 | 5 | 0 | 0
Not completed — Lost to Follow-up | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Protocol Deviation | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Not completed — Withdrawal by Subject | 4 | 2 | 1 | 0 | 0 | 0 | 0 | 1 | 2
Not completed — Other | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- FE 201836 500 µg (Randomized Treatment Period): FE 201836 500 µg oral solution and placebo ODT, administered once daily
- Desmopressin 25µg (Randomized Treatment Period): Desmopressin 25 µg ODT and placebo oral solution, administered once daily (female subjects)
- Total: Total of all reporting groups
Arm/Group | FE 201836 500 µg (Randomized Treatment Period) | FE 201836 350 µg (Randomized Treatment Period) | FE 201836 250 µg (Randomized Treatment Period) | FE 201836 150 µg (Randomized Treatment Period) | FE 201836 100 µg (Randomized Treatment Period) | FE 201836 50 µg (Randomized Treatment Period) | Placebo (Randomized Treatment Period) | Desmopressin 25µg (Randomized Treatment Period) | Desmopressin 50 µg (Randomized Treatment Period) | Total
Number analyzed (Participants) | 60 | 27 | 24 | 14 | 13 | 34 | 87 | 26 | 17 | 302
Age, Continuous [Mean (Standard Deviation); unit: years] | 59.0 (14.1) | 58.0 (14.3) | 60.8 (13.0) | 63.9 (7.5) | 61.5 (9.2) | 59.1 (10.4) | 58.9 (13.9) | 51.1 (11.1) | 60.9 (9.5) | 58.8 (12.8)
Age, Customized [Number; unit: years]
  <65 years old | 35 | 19 | 14 | 6 | 6 | 21 | 52 | 24 | 11 | 188
  >=65 years old | 25 | 8 | 10 | 8 | 7 | 13 | 35 | 2 | 6 | 114
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 40 | 18 | 16 | 5 | 8 | 16 | 51 | 26 | 0 | 180
  Male | 20 | 9 | 8 | 9 | 5 | 18 | 36 | 0 | 17 | 122
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants] — Population: Number analyzed differs from the overall population as baseline ethnicity was not reported for some of the subjects.
  Participants
    number analyzed (Participants) | 59 | 27 | 24 | 14 | 13 | 34 | 86 | 26 | 17 | 300
    Hispanic or Latino | 17 | 9 | 6 | 3 | 7 | 12 | 35 | 12 | 4 | 105
    Not Hispanic or Latino | 42 | 18 | 18 | 11 | 6 | 22 | 51 | 14 | 13 | 195
    Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants] — Population: Number analyzed differs from the overall population as baseline race was not reported for some of the subjects.
  Participants
    number analyzed (Participants) | 60 | 27 | 24 | 14 | 13 | 33 | 86 | 26 | 17 | 300
    American Indian or Alaska Native | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 0 | 0 | 3
    Asian | 2 | 0 | 0 | 0 | 0 | 0 | 2 | 1 | 0 | 5
    Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
    Black or African American | 6 | 3 | 2 | 0 | 1 | 1 | 5 | 6 | 4 | 28
    White | 52 | 24 | 22 | 14 | 11 | 31 | 78 | 19 | 13 | 264
    More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
    Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Baseline body mass index (BMI) [Mean (Standard Deviation); unit: kg/m^2] | 30.66 (6.05) | 29.91 (4.64) | 29.56 (6.50) | 32.03 (8.26) | 31.52 (4.60) | 30.93 (6.16) | 29.54 (5.14) | 31.89 (7.99) | 31.05 (6.49) | 30.44 (6.00)
Mean Number of Nocturnal Voids [Mean (Standard Deviation); unit: nocturnal voids] — Population: Number analyzed differs from the overall population as baseline mean number of nocturnal voids was not calculated for some of the subjects.
  nocturnal voids
    number analyzed (Participants) | 59 | 27 | 24 | 14 | 13 | 34 | 86 | 25 | 17 | 299
    (all) | 2.88 (0.84) | 3.01 (0.72) | 3.10 (1.11) | 2.98 (0.84) | 3.33 (0.82) | 3.24 (1.18) | 3.09 (0.83) | 3.38 (1.45) | 3.16 (1.22) | 3.09 (0.98)
Mean Nocturnal Urine Volume (NUV) [Mean (Standard Deviation); unit: mL] — Population: Number analyzed differs from the overall population as baseline mean NUV was not calculated for some of the subjects.
  mL
    number analyzed (Participants) | 58 | 26 | 24 | 14 | 13 | 34 | 86 | 25 | 17 | 297
    (all) | 804.6 (313.8) | 766.0 (242.1) | 897.3 (373.6) | 803.1 (304.7) | 892.4 (206.7) | 879.9 (354.1) | 752.3 (269.5) | 839.3 (286.4) | 803.5 (425.8) | 808.8 (307.5)
Mean Nocturnal Polyuria Index [Mean (Standard Deviation); unit: percentage] — Nocturnal polyuria index (NPi) is calculated by dividing the nocturnal urine volume (NUV) by the 24-hour urine volume. In this clinical trial the NPi definition >33% is used for all ages to define presence of nocturnal polyuria (NP). Population: Number analyzed differs from the overall population as baseline mean nocturnal polyuria index was not calculated for some of the subjects.
  percentage
    number analyzed (Participants) | 55 | 25 | 22 | 14 | 12 | 31 | 76 | 23 | 16 | 274
    (all) | 48.87 (12.04) | 46.76 (10.08) | 49.75 (15.96) | 50.99 (12.93) | 44.59 (6.58) | 47.01 (9.86) | 47.91 (14.29) | 49.21 (13.93) | 49.10 (17.93) | 48.24 (12.99)
Mean Nocturia Impact (NI) Diary Total Score [Mean (Standard Deviation); unit: score on a scale] — Population: Number analyzed differs from the overall population as mean NI Diary Total Score was not calculated for some of the subjects.
  score on a scale
    number analyzed (Participants) | 60 | 26 | 24 | 14 | 13 | 32 | 86 | 25 | 17 | 297
    (all) | 47.20 (18.39) | 47.03 (28.44) | 38.76 (19.09) | 36.28 (22.10) | 51.63 (17.73) | 42.46 (23.28) | 47.66 (21.25) | 58.06 (20.78) | 39.88 (23.08) | 46.30 (21.81)
Mean NI Diary Overall Impact Score [Mean (Standard Deviation); unit: score on a scale] — The Nocturia Impact (NI) Diary is a 12-item questionnaire with 11 core items (Q1-Q11) and an overall Quality-of-Life (QoL) impact question (Q12). For the overall impact question (Q12), response options range from 0 (not at all) to 4 (a great deal). The NI Diary Overall Impact Score is standardized from 0 to 100 (lowest to highest impact). The score at each visit was calculated as the average over the three consecutive 24-hour periods just prior to the respective visit. Population: Number analyzed differs from the overall population as mean NI Diary Overall Impact Score was not calculated for some of the subjects.
  score on a scale
    number analyzed (Participants) | 60 | 26 | 24 | 14 | 13 | 32 | 86 | 25 | 17 | 297
    (all) | 59.2 (25.4) | 62.3 (29.8) | 55.9 (21.6) | 53.0 (30.6) | 68.6 (20.7) | 59.9 (26.8) | 62.7 (26.8) | 71.5 (23.8) | 54.2 (28.0) | 61.2 (26.3)
Insomnia Severity Index (ISI) [Mean (Standard Deviation); unit: score on a scale] — The Insomnia Severity Index (ISI) is a 7-item questionnaire which comprises of four 'sleep-related' items and three 'wake-related' items. Each item is rated on a 0-4 scale and the total score ranges from 0 to 28 (higher score suggests more severe insomnia). Population: Number analyzed differs from the overall population as mean ISI was not calculated for some of the subjects.
  score on a scale
    number analyzed (Participants) | 55 | 26 | 24 | 14 | 9 | 31 | 77 | 26 | 17 | 279
    (all) | 15.8 (5.4) | 15.7 (6.1) | 14.3 (5.1) | 13.0 (6.7) | 16.4 (5.6) | 14.7 (4.8) | 15.6 (5.8) | 18.2 (4.7) | 15.5 (6.8) | 15.6 (5.6)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Aggregated Mean Number of Nocturnal Voids During 12 Weeks of Treatment
Description: Nocturnal voids were defined as voids occuring from 5 minutes after bedtime until rising in the morning.
  The number of nocturnal voids at each visit was calculated as the average over the 3 consecutive 24 hour periods just prior to the respective visit. The visit-specific means were aggregated into a mean of current and preceding visits.
  Level estimated for baseline value of mean number of nocturnal voids equal to 2, and 95% credibility interval (2.5 and 97.5 percentiles of the posterior distribution) instead of confidence interval are presented in this endpoint.
Time Frame: Baseline, during 12 weeks of treatment
Population: The intention-to-treat analysis set for the randomized treatment period (ITT-RT) comprised of all the subjects randomized at Visit 4.
Measure: Mean (95% Confidence Interval); unit: nocturnal voids
Groups:
- FE 201836 500 ug (Randomized Treatment Period): FE 201836 500 µg oral solution and placebo ODT, administered once daily
- FE 201836 350 ug (Randomized Treatment Period): FE 201836 350 µg oral solution and placebo ODT, administered once daily
- FE 201836 250 ug (Randomized Treatment Period): FE 201836 250 µg oral solution and placebo ODT, administered once daily
- FE 201836 150 ug (Randomized Treatment Period): FE 201836 150 µg oral solution and placebo ODT, administered once daily
- FE 201836 100 ug (Randomized Treatment Period): FE 201836 100 µg oral solution and placebo ODT, administered once daily
- FE 201836 50 ug (Randomized Treatment Period): FE 201836 50 µg oral solution and placebo ODT, administered once daily
Arm/Group | FE 201836 500 ug (Randomized Treatment Period) | FE 201836 350 ug (Randomized Treatment Period) | FE 201836 250 ug (Randomized Treatment Period) | FE 201836 150 ug (Randomized Treatment Period) | FE 201836 100 ug (Randomized Treatment Period) | FE 201836 50 ug (Randomized Treatment Period) | Placebo (Randomized Treatment Period)
Number analyzed (Participants) | 60 | 27 | 24 | 14 | 13 | 34 | 87
nocturnal voids | -1.06 [-1.28 to -0.86] | -0.99 [-1.20 to -0.78] | -0.89 [-1.12 to -0.69] | -0.80 [-1.00 to -0.62] | -0.77 [-0.97 to -0.59] | -0.76 [-0.95 to -0.58] | -0.76 [-0.95 to -0.58]
Statistical Analysis 1: Comparison: FE 201836 500 ug (Randomized Treatment Period) vs Placebo (Randomized Treatment Period); Based on a Bayesian analysis of a sigmoidal dose-response relationship; Test type: Superiority; Mean Difference = -0.30, 95% CI 2-sided [-0.54 to -0.07]
Statistical Analysis 2: Comparison: FE 201836 350 ug (Randomized Treatment Period) vs Placebo (Randomized Treatment Period); Based on a Bayesian analysis of a sigmoidal dose-response relationship; Test type: Superiority; Mean Difference = -0.23, 95% CI 2-sided [-0.46 to -0.02]
Statistical Analysis 3: Comparison: FE 201836 250 ug (Randomized Treatment Period) vs Placebo (Randomized Treatment Period); Based on a Bayesian analysis of a sigmoidal dose-response relationship; Test type: Superiority; Mean Difference = -0.14, 95% CI 2-sided [-0.36 to -0.00]
Statistical Analysis 4: Comparison: FE 201836 150 ug (Randomized Treatment Period) vs Placebo (Randomized Treatment Period); Based on a Bayesian analysis of a sigmoidal dose-response relationship; Test type: Superiority; Mean Difference = -0.040, 95% CI 2-sided [-0.23 to -0.00]
Statistical Analysis 5: Comparison: FE 201836 100 ug (Randomized Treatment Period) vs Placebo (Randomized Treatment Period); Based on a Bayesian analysis of a sigmoidal dose-response relationship; Test type: Superiority; Mean Difference = -0.02, 95% CI 2-sided [-0.14 to -0.00]
Statistical Analysis 6: Comparison: FE 201836 50 ug (Randomized Treatment Period) vs Placebo (Randomized Treatment Period); Based on a Bayesian analysis of a sigmoidal dose-response relationship; Test type: Superiority; Mean Difference = -0.01, 95% CI 2-sided [-0.07 to -0.00]

2. Secondary Outcome: Change From Baseline in Mean Number of Nocturnal Voids at Week 1
Description: Nocturnal voids were defined as voids occuring from 5 minutes after bedtime until rising in the morning.
  The number of nocturnal voids at each visit was calculated as the average over the 3 consecutive 24 hour periods just prior to the respective visit. Adjusted visit-specific mean changes from baseline in nocturnal voids are estimated using a baseline value of 2.
  MMRM=Mixed Model for Repeated Measurements.
  For all visit-specific results, the tables present the number of subjects with an observation of the endpoints in question at the specific visit. All secondary analyses are performed using the observed-case approach based on repeated measurements for all subjects in the ITT-RT population. That is, these secondary analyses are based on all subjects with at least one non-missing post-baseline observation (with a baseline value if relevant).
Time Frame: Baseline, Week 1
Population: The ITT-RT comprised of all the subjects randomized at Visit 4.
Measure: Mean (95% Confidence Interval); unit: nocturnal voids
Arm/Group | FE 201836 500 ug (Randomized Treatment Period) | FE 201836 350 ug (Randomized Treatment Period) | FE 201836 250 ug (Randomized Treatment Period) | FE 201836 150 ug (Randomized Treatment Period) | FE 201836 100 ug (Randomized Treatment Period) | FE 201836 50 ug (Randomized Treatment Period) | Placebo (Randomized Treatment Period)
Number analyzed (Participants) | 54 | 24 | 24 | 14 | 11 | 33 | 80
nocturnal voids | -0.714 [-1.005 to -0.424] | -1.162 [-1.577 to -0.747] | -0.722 [-1.149 to -0.296] | -0.520 [-1.058 to 0.017] | -0.722 [-1.318 to -0.126] | -0.325 [-0.709 to 0.059] | -0.575 [-0.842 to -0.308]
Statistical Analysis 1: Comparison: FE 201836 500 ug (Randomized Treatment Period) vs Placebo (Randomized Treatment Period); Test type: Superiority; p = 0.4214, MMRM — Threshold for significance at 0.05 level; Mean Difference = -0.139, 95% CI 2-sided [-0.480 to 0.201]
Statistical Analysis 2: Comparison: FE 201836 350 ug (Randomized Treatment Period) vs Placebo (Randomized Treatment Period); Test type: Superiority; p = 0.0101, MMRM — Threshold for significance at 0.05 level; Mean Difference = -0.587, 95% CI 2-sided [-1.034 to -0.141]
Statistical Analysis 3: Comparison: FE 201836 250 ug (Randomized Treatment Period) vs Placebo (Randomized Treatment Period); Test type: Superiority; p = 0.5203, MMRM — Threshold for significance at 0.05 level; Mean Difference = -0.148, 95% CI 2-sided [-0.599 to 0.304]
Statistical Analysis 4: Comparison: FE 201836 150 ug (Randomized Treatment Period) vs Placebo (Randomized Treatment Period); Test type: Superiority; p = 0.8483, MMRM — Threshold for significance at 0.05 level; Mean Difference = 0.055, 95% CI 2-sided [-0.508 to 0.617]
Statistical Analysis 5: Comparison: FE 201836 100 ug (Randomized Treatment Period) vs Placebo (Randomized Treatment Period); Test type: Superiority; p = 0.6357, MMRM — Threshold for significance at 0.05 level; Mean Difference = -0.147, 95% CI 2-sided [-0.759 to 0.464]
Statistical Analysis 6: Comparison: FE 201836 50 ug (Randomized Treatment Period) vs Placebo (Randomized Treatment Period); Test type: Superiority; p = 0.2222, MMRM — Threshold for significance at 0.05 level; Mean Difference = 0.250, 95% CI 2-sided [-0.152 to 0.652]

3. Secondary Outcome: Change From Baseline in Mean Number of Nocturnal Voids at Week 4
Description: Nocturnal voids were defined as voids occuring from 5 minutes after bedtime until rising in the morning.
  The number of nocturnal voids at each visit was calculated as the average over the 3 consecutive 24 hour periods just prior to the respective visit. Adjusted visit-specific mean changes from baseline in nocturnal voids are estimated using a baseline value of 2.
Time Frame: Baseline, Week 4
Population: The ITT-RT comprised of all the subjects randomized at Visit 4.
Measure: Mean (95% Confidence Interval); unit: nocturnal voids
Arm/Group | FE 201836 500 ug (Randomized Treatment Period) | FE 201836 350 ug (Randomized Treatment Period) | FE 201836 250 ug (Randomized Treatment Period) | FE 201836 150 ug (Randomized Treatment Period) | FE 201836 100 ug (Randomized Treatment Period) | FE 201836 50 ug (Randomized Treatment Period) | Placebo (Randomized Treatment Period)
Number analyzed (Participants) | 50 | 22 | 21 | 12 | 12 | 31 | 76
nocturnal voids | -1.078 [-1.345 to -0.811] | -1.330 [-1.708 to -0.952] | -0.784 [-1.181 to -0.386] | -0.471 [-0.969 to 0.028] | -0.952 [-1.469 to -0.435] | -0.518 [-0.866 to -0.171] | -0.912 [-1.152 to -0.673]
Statistical Analysis 1: Comparison: FE 201836 500 ug (Randomized Treatment Period) vs Placebo (Randomized Treatment Period); Test type: Superiority; p = 0.2909, MMRM — Threshold for significance at 0.05 level; Mean Difference = -0.166, 95% CI 2-sided [-0.474 to 0.143]
Statistical Analysis 2: Comparison: FE 201836 350 ug (Randomized Treatment Period) vs Placebo (Randomized Treatment Period); Test type: Superiority; p = 0.0440, MMRM — Threshold for significance at 0.05 level; Mean Difference = -0.418, 95% CI 2-sided [-0.824 to -0.011]
Statistical Analysis 3: Comparison: FE 201836 250 ug (Randomized Treatment Period) vs Placebo (Randomized Treatment Period); Test type: Superiority; p = 0.5438, MMRM — Threshold for significance at 0.05 level; Mean Difference = 0.128, 95% CI 2-sided [-0.288 to 0.545]
Statistical Analysis 4: Comparison: FE 201836 150 ug (Randomized Treatment Period) vs Placebo (Randomized Treatment Period); Test type: Superiority; p = 0.0960, MMRM — Threshold for significance at 0.05 level; Mean Difference = 0.441, 95% CI 2-sided [-0.079 to 0.962]
Statistical Analysis 5: Comparison: FE 201836 100 ug (Randomized Treatment Period) vs Placebo (Randomized Treatment Period); Test type: Superiority; p = 0.8826, MMRM — Threshold for significance at 0.05 level; Mean Difference = -0.040, 95% CI 2-sided [-0.568 to 0.488]
Statistical Analysis 6: Comparison: FE 201836 50 ug (Randomized Treatment Period) vs Placebo (Randomized Treatment Period); Test type: Superiority; p = 0.0344, MMRM — Threshold for significance at 0.05 level; Mean Difference = 0.394, 95% CI 2-sided [0.029 to 0.759]

4. Secondary Outcome: Change From Baseline in Mean Number of Nocturnal Voids at Week 8
Description: as for outcome 3
Time Frame: Baseline, Week 8
Population: The ITT-RT comprised of all the subjects randomized at Visit 4.
Measure: Mean (95% Confidence Interval); unit: nocturnal voids
Arm/Group | FE 201836 500 ug (Randomized Treatment Period) | FE 201836 350 ug (Randomized Treatment Period) | FE 201836 250 ug (Randomized Treatment Period) | FE 201836 150 ug (Randomized Treatment Period) | FE 201836 100 ug (Randomized Treatment Period) | FE 201836 50 ug (Randomized Treatment Period) | Placebo (Randomized Treatment Period)
Number analyzed (Participants) | 44 | 23 | 21 | 14 | 12 | 30 | 70
nocturnal voids | -1.085 [-1.394 to -0.776] | -1.177 [-1.603 to -0.751] | -0.965 [-1.414 to -0.516] | -0.490 [-1.037 to 0.058] | -1.077 [-1.671 to -0.484] | -0.786 [-1.187 to -0.386] | -0.953 [-1.233 to -0.672]
Statistical Analysis 1: Comparison: FE 201836 500 ug (Randomized Treatment Period) vs Placebo (Randomized Treatment Period); Test type: Superiority; p = 0.4732, MMRM — Threshold for significance at 0.05 level; Mean Difference = -0.132, 95% CI 2-sided [-0.496 to 0.231]
Statistical Analysis 2: Comparison: FE 201836 350 ug (Randomized Treatment Period) vs Placebo (Randomized Treatment Period); Test type: Superiority; p = 0.3394, MMRM — Threshold for significance at 0.05 level; Mean Difference = -0.224, 95% CI 2-sided [-0.685 to 0.237]
Statistical Analysis 3: Comparison: FE 201836 250 ug (Randomized Treatment Period) vs Placebo (Randomized Treatment Period); Test type: Superiority; p = 0.9600, MMRM — Threshold for significance at 0.05 level; Mean Difference = -0.012, 95% CI 2-sided [-0.488 to 0.463]
Statistical Analysis 4: Comparison: FE 201836 150 ug (Randomized Treatment Period) vs Placebo (Randomized Treatment Period); Test type: Superiority; p = 0.1131, MMRM — Threshold for significance at 0.05 level; Mean Difference = 0.463, 95% CI 2-sided [-0.111 to 1.037]
Statistical Analysis 5: Comparison: FE 201836 100 ug (Randomized Treatment Period) vs Placebo (Randomized Treatment Period); Test type: Superiority; p = 0.6853, MMRM — Threshold for significance at 0.05 level; Mean Difference = -0.124, 95% CI 2-sided [-0.729 to 0.480]
Statistical Analysis 6: Comparison: FE 201836 50 ug (Randomized Treatment Period) vs Placebo (Randomized Treatment Period); Test type: Superiority; p = 0.4364, MMRM — Threshold for significance at 0.05 level; Mean Difference = 0.166, 95% CI 2-sided [-0.254 to 0.587]

5. Secondary Outcome: Change From Baseline in Mean Number of Nocturnal Voids at Week 12
Description: as for outcome 3
Time Frame: Baseline, Week 12
Population: The ITT-RT comprised of all the subjects randomized at Visit 4.
Measure: Mean (95% Confidence Interval); unit: nocturnal voids
Arm/Group | FE 201836 500 ug (Randomized Treatment Period) | FE 201836 350 ug (Randomized Treatment Period) | FE 201836 250 ug (Randomized Treatment Period) | FE 201836 150 ug (Randomized Treatment Period) | FE 201836 100 ug (Randomized Treatment Period) | FE 201836 50 ug (Randomized Treatment Period) | Placebo (Randomized Treatment Period)
Number analyzed (Participants) | 40 | 19 | 19 | 14 | 11 | 29 | 69
nocturnal voids | -1.256 [-1.568 to -0.944] | -1.120 [-1.558 to -0.683] | -0.850 [-1.301 to -0.400] | -0.674 [-1.206 to -0.142] | -1.053 [-1.650 to -0.456] | -0.921 [-1.317 to -0.524] | -0.957 [-1.237 to -0.677]
Statistical Analysis 1: Comparison: FE 201836 500 ug (Randomized Treatment Period) vs Placebo (Randomized Treatment Period); Test type: Superiority; p = 0.1106, MMRM — Threshold for significance at 0.05 level; Mean Difference = -0.299, 95% CI 2-sided [-0.667 to 0.069]
Statistical Analysis 2: Comparison: FE 201836 350 ug (Randomized Treatment Period) vs Placebo (Randomized Treatment Period); Test type: Superiority; p = 0.5005, MMRM — Threshold for significance at 0.05 level; Mean Difference = -0.163, 95% CI 2-sided [-0.639 to 0.313]
Statistical Analysis 3: Comparison: FE 201836 250 ug (Randomized Treatment Period) vs Placebo (Randomized Treatment Period); Test type: Superiority; p = 0.6604, MMRM — Threshold for significance at 0.05 level; Mean Difference = 0.107, 95% CI 2-sided [-0.372 to 0.586]
Statistical Analysis 4: Comparison: FE 201836 150 ug (Randomized Treatment Period) vs Placebo (Randomized Treatment Period); Test type: Superiority; p = 0.3178, MMRM — Threshold for significance at 0.05 level; Mean Difference = 0.283, 95% CI 2-sided [-0.275 to 0.842]
Statistical Analysis 5: Comparison: FE 201836 100 ug (Randomized Treatment Period) vs Placebo (Randomized Treatment Period); Test type: Superiority; p = 0.7561, MMRM — Threshold for significance at 0.05 level; Mean Difference = -0.096, 95% CI 2-sided [-0.701 to 0.510]
Statistical Analysis 6: Comparison: FE 201836 50 ug (Randomized Treatment Period) vs Placebo (Randomized Treatment Period); Test type: Superiority; p = 0.8614, MMRM — Threshold for significance at 0.05 level; Mean Difference = 0.037, 95% CI 2-sided [-0.378 to 0.452]

6. Secondary Outcome: Responder Rate in Nocturnal Voids at Week 1
Description: Defined as 50% reduction in nocturnal voids from baseline.
  Adjusted visit-specific estimated odds of at least 50% in the reduction mean number of nocturnal voids are estimated using a baseline value of 2.
  The estimated odd equals the probability of response divided by the probability of non-response; these odds may vary between 0 and infinity. For example, if the probability of responding is 80%, the odd of responding is 4, as it is 4 times more likely to respond (80%) then it is not to respond (20%).
Time Frame: Week 1
Population: The ITT-RT comprised of all the subjects randomized at Visit 4.
Measure: Mean (95% Confidence Interval); unit: odd of response
Arm/Group | FE 201836 500 ug (Randomized Treatment Period) | FE 201836 350 ug (Randomized Treatment Period) | FE 201836 250 ug (Randomized Treatment Period) | FE 201836 150 ug (Randomized Treatment Period) | FE 201836 100 ug (Randomized Treatment Period) | FE 201836 50 ug (Randomized Treatment Period) | Placebo (Randomized Treatment Period)
Number analyzed (Participants) | 54 | 24 | 24 | 14 | 11 | 33 | 80
odd of response | 0.844 [0.457 to 1.558] | 1.202 [0.510 to 2.833] | 0.682 [0.280 to 1.662] | 0.818 [0.269 to 2.490] | 0.810 [0.240 to 2.738] | 0.513 [0.227 to 1.157] | 0.480 [0.272 to 0.848]
Statistical Analysis 1: Comparison: FE 201836 500 ug (Randomized Treatment Period) vs Placebo (Randomized Treatment Period); Test type: Superiority; p = 0.117, Regression, Logistic — Threshold for significance at 0.05 level; Odds Ratio (OR) = 1.759, 95% CI 2-sided [0.869 to 3.560]
Statistical Analysis 2: Comparison: FE 201836 350 ug (Randomized Treatment Period) vs Placebo (Randomized Treatment Period); Test type: Superiority; p = 0.048, Regression, Logistic — Threshold for significance at 0.05 level; Odds Ratio (OR) = 2.505, 95% CI 2-sided [1.010 to 6.214]
Statistical Analysis 3: Comparison: FE 201836 250 ug (Randomized Treatment Period) vs Placebo (Randomized Treatment Period); Test type: Superiority; p = 0.460, Regression, Logistic — Threshold for significance at 0.05 level; Odds Ratio (OR) = 1.420, 95% CI 2-sided [0.560 to 3.602]
Statistical Analysis 4: Comparison: FE 201836 150 ug (Randomized Treatment Period) vs Placebo (Randomized Treatment Period); Test type: Superiority; p = 0.367, Regression, Logistic — Threshold for significance at 0.05 level; Odds Ratio (OR) = 1.704, 95% CI 2-sided [0.535 to 5.427]
Statistical Analysis 5: Comparison: FE 201836 100 ug (Randomized Treatment Period) vs Placebo (Randomized Treatment Period); Test type: Superiority; p = 0.407, Regression, Logistic — Threshold for significance at 0.05 level; Odds Ratio (OR) = 1.689, 95% CI 2-sided [0.489 to 5.825]
Statistical Analysis 6: Comparison: FE 201836 50 ug (Randomized Treatment Period) vs Placebo (Randomized Treatment Period); Test type: Superiority; p = 0.876, Regression, Logistic — Threshold for significance at 0.05 level; Odds Ratio (OR) = 1.069, 95% CI 2-sided [0.462 to 2.473]

7. Secondary Outcome: Responder Rate in Nocturnal Voids at Week 4
Description: Defined as 50% reduction in nocturnal voids from baseline.
  Adjusted visit-specific estimated odds of at least 50% reduction in the mean number of nocturnal voids are estimated using a baseline value of 2.
  The estimated odd equals the probability of response divided by the probability of non-response; these odds may vary between 0 and infinity. For example, if the probability of responding is 80%, the odd of responding is 4, as it is 4 times more likely to respond (80%) then it is not to respond (20%).
Time Frame: Week 4
Population: The ITT-RT comprised of all the subjects randomized at Visit 4.
Measure: Mean (95% Confidence Interval); unit: odd of response
Arm/Group | FE 201836 500 ug (Randomized Treatment Period) | FE 201836 350 ug (Randomized Treatment Period) | FE 201836 250 ug (Randomized Treatment Period) | FE 201836 150 ug (Randomized Treatment Period) | FE 201836 100 ug (Randomized Treatment Period) | FE 201836 50 ug (Randomized Treatment Period) | Placebo (Randomized Treatment Period)
Number analyzed (Participants) | 50 | 22 | 21 | 12 | 12 | 31 | 76
odd of response | 1.199 [0.633 to 2.270] | 5.851 [1.511 to 22.650] | 0.634 [0.255 to 1.575] | 0.534 [0.165 to 1.731] | 1.760 [0.470 to 6.596] | 0.683 [0.301 to 1.550] | 1.235 [0.686 to 2.224]
Statistical Analysis 1: Comparison: FE 201836 500 ug (Randomized Treatment Period) vs Placebo (Randomized Treatment Period); Test type: Superiority; p = 0.937, Regression, Logistic — Threshold for significance at 0.05 level; Odds Ratio (OR) = 0.971, 95% CI 2-sided [0.470 to 2.005]
Statistical Analysis 2: Comparison: FE 201836 350 ug (Randomized Treatment Period) vs Placebo (Randomized Treatment Period); Test type: Superiority; p = 0.028, Regression, Logistic — Threshold for significance at 0.05 level; Odds Ratio (OR) = 4.738, 95% CI 2-sided [1.183 to 18.968]
Statistical Analysis 3: Comparison: FE 201836 250 ug (Randomized Treatment Period) vs Placebo (Randomized Treatment Period); Test type: Superiority; p = 0.166, Regression, Logistic — Threshold for significance at 0.05 level; Odds Ratio (OR) = 0.513, 95% CI 2-sided [0.200 to 1.318]
Statistical Analysis 4: Comparison: FE 201836 150 ug (Randomized Treatment Period) vs Placebo (Randomized Treatment Period); Test type: Superiority; p = 0.174, Regression, Logistic — Threshold for significance at 0.05 level; Odds Ratio (OR) = 0.433, 95% CI 2-sided [0.129 to 1.447]
Statistical Analysis 5: Comparison: FE 201836 100 ug (Randomized Treatment Period) vs Placebo (Randomized Treatment Period); Test type: Superiority; p = 0.608, Regression, Logistic — Threshold for significance at 0.05 level; Odds Ratio (OR) = 1.425, 95% CI 2-sided [0.369 to 5.512]
Statistical Analysis 6: Comparison: FE 201836 50 ug (Randomized Treatment Period) vs Placebo (Randomized Treatment Period); Test type: Superiority; p = 0.171, Regression, Logistic — Threshold for significance at 0.05 level; Odds Ratio (OR) = 0.553, 95% CI 2-sided [0.237 to 1.292]

8. Secondary Outcome: Responder Rate in Nocturnal Voids at Week 8
Description: as for outcome 7
Time Frame: Week 8
Population: The ITT-RT comprised of all the subjects randomized at Visit 4.
Measure: Mean (95% Confidence Interval); unit: odd of response
Arm/Group | FE 201836 500 ug (Randomized Treatment Period) | FE 201836 350 ug (Randomized Treatment Period) | FE 201836 250 ug (Randomized Treatment Period) | FE 201836 150 ug (Randomized Treatment Period) | FE 201836 100 ug (Randomized Treatment Period) | FE 201836 50 ug (Randomized Treatment Period) | Placebo (Randomized Treatment Period)
Number analyzed (Participants) | 44 | 23 | 21 | 14 | 12 | 30 | 70
odd of response | 1.395 [0.717 to 2.715] | 3.398 [1.150 to 10.043] | 1.928 [0.721 to 5.155] | 0.877 [0.286 to 2.688] | 1.039 [0.302 to 3.569] | 1.489 [0.638 to 3.474] | 1.503 [0.806 to 2.803]
Statistical Analysis 1: Comparison: FE 201836 500 ug (Randomized Treatment Period) vs Placebo (Randomized Treatment Period); Test type: Superiority; p = 0.850, Regression, Logistic — Threshold for significance at 0.05 level; Odds Ratio (OR) = 0.928, 95% CI 2-sided [0.430 to 2.003]
Statistical Analysis 2: Comparison: FE 201836 350 ug (Randomized Treatment Period) vs Placebo (Randomized Treatment Period); Test type: Superiority; p = 0.150, Regression, Logistic — Threshold for significance at 0.05 level; Odds Ratio (OR) = 2.261, 95% CI 2-sided [0.745 to 6.862]
Statistical Analysis 3: Comparison: FE 201836 250 ug (Randomized Treatment Period) vs Placebo (Randomized Treatment Period); Test type: Superiority; p = 0.632, Regression, Logistic — Threshold for significance at 0.05 level; Odds Ratio (OR) = 1.283, 95% CI 2-sided [0.462 to 3.566]
Statistical Analysis 4: Comparison: FE 201836 150 ug (Randomized Treatment Period) vs Placebo (Randomized Treatment Period); Test type: Superiority; p = 0.363, Regression, Logistic — Threshold for significance at 0.05 level; Odds Ratio (OR) = 0.583, 95% CI 2-sided [0.183 to 1.863]
Statistical Analysis 5: Comparison: FE 201836 100 ug (Randomized Treatment Period) vs Placebo (Randomized Treatment Period); Test type: Superiority; p = 0.555, Regression, Logistic — Threshold for significance at 0.05 level; Odds Ratio (OR) = 0.691, 95% CI 2-sided [0.203 to 2.359]
Statistical Analysis 6: Comparison: FE 201836 50 ug (Randomized Treatment Period) vs Placebo (Randomized Treatment Period); Test type: Superiority; p = 0.984, Regression, Logistic — Threshold for significance at 0.05 level; Odds Ratio (OR) = 0.991, 95% CI 2-sided [0.408 to 2.405]

9. Secondary Outcome: Responder Rate in Nocturnal Voids at Week 12
Description: as for outcome 7
Time Frame: Week 12
Population: The ITT-RT comprised of all the subjects randomized at Visit 4.
Measure: Mean (95% Confidence Interval); unit: odd of response
Arm/Group | FE 201836 500 ug (Randomized Treatment Period) | FE 201836 350 ug (Randomized Treatment Period) | FE 201836 250 ug (Randomized Treatment Period) | FE 201836 150 ug (Randomized Treatment Period) | FE 201836 100 ug (Randomized Treatment Period) | FE 201836 50 ug (Randomized Treatment Period) | Placebo (Randomized Treatment Period)
Number analyzed (Participants) | 40 | 19 | 19 | 14 | 11 | 29 | 69
odd of response | 3.914 [1.830 to 8.370] | 1.891 [0.693 to 5.163] | 1.824 [0.694 to 4.795] | 0.854 [0.279 to 2.611] | 1.400 [0.401 to 4.893] | 1.395 [0.611 to 3.181] | 1.590 [0.844 to 2.993]
Statistical Analysis 1: Comparison: FE 201836 500 ug (Randomized Treatment Period) vs Placebo (Randomized Treatment Period); Test type: Superiority; p = 0.046, Regression, Logistic — Threshold for significance at 0.05 level; Odds Ratio (OR) = 2.462, 95% CI 2-sided [1.017 to 5.961]
Statistical Analysis 2: Comparison: FE 201836 350 ug (Randomized Treatment Period) vs Placebo (Randomized Treatment Period); Test type: Superiority; p = 0.745, Regression, Logistic — Threshold for significance at 0.05 level; Odds Ratio (OR) = 1.190, 95% CI 2-sided [0.418 to 3.386]
Statistical Analysis 3: Comparison: FE 201836 250 ug (Randomized Treatment Period) vs Placebo (Randomized Treatment Period); Test type: Superiority; p = 0.790, Regression, Logistic — Threshold for significance at 0.05 level; Odds Ratio (OR) = 1.147, 95% CI 2-sided [0.417 to 3.155]
Statistical Analysis 4: Comparison: FE 201836 150 ug (Randomized Treatment Period) vs Placebo (Randomized Treatment Period); Test type: Superiority; p = 0.293, Regression, Logistic — Threshold for significance at 0.05 level; Odds Ratio (OR) = 0.537, 95% CI 2-sided [0.169 to 1.710]
Statistical Analysis 5: Comparison: FE 201836 100 ug (Randomized Treatment Period) vs Placebo (Randomized Treatment Period); Test type: Superiority; p = 0.843, Regression, Logistic — Threshold for significance at 0.05 level; Odds Ratio (OR) = 0.881, 95% CI 2-sided [0.252 to 3.076]
Statistical Analysis 6: Comparison: FE 201836 50 ug (Randomized Treatment Period) vs Placebo (Randomized Treatment Period); Test type: Superiority; p = 0.763, Regression, Logistic — Threshold for significance at 0.05 level; Odds Ratio (OR) = 0.877, 95% CI 2-sided [0.375 to 2.053]

10. Secondary Outcome: Responder Rate in Nocturnal Voids During 12 Weeks of Treatment
Description: Defined as 50% reduction in nocturnal voids from baseline.
  Estimated odds of at least 50% reduction in the aggregated mean number of nocturnal voids for a subject with 2 nocturnal voids at baseline are presented in this endpoint.
  The 95% credibility interval (2.5 and 97.5 percentiles of the posterior distribution) instead of confidence interval is presented for this endpoint.
  The estimated odd equals the probability of response divided by the probability of non-response; these odds may vary between 0 and infinity. For example, if the probability of responding is 80%, the odd of responding is 4, as it is 4 times more likely to respond (80%) then it is not to respond (20%).
Time Frame: During 12 weeks of treatment
Population: The ITT-RT comprised of all the subjects randomized at Visit 4.
Measure: Mean (95% Confidence Interval); unit: odd of response
Arm/Group | FE 201836 500 ug (Randomized Treatment Period) | FE 201836 350 ug (Randomized Treatment Period) | FE 201836 250 ug (Randomized Treatment Period) | FE 201836 150 ug (Randomized Treatment Period) | FE 201836 100 ug (Randomized Treatment Period) | FE 201836 50 ug (Randomized Treatment Period) | Placebo (Randomized Treatment Period)
Number analyzed (Participants) | 60 | 27 | 24 | 14 | 13 | 34 | 87
odd of response | 1.129 [0.808 to 1.753] | 1.095 [0.772 to 1.661] | 1.032 [0.711 to 1.543] | 0.934 [0.597 to 1.378] | 0.887 [0.555 to 1.253] | 0.849 [0.534 to 1.187] | 0.834 [0.514 to 1.180]
Statistical Analysis 1: Comparison: FE 201836 500 ug (Randomized Treatment Period) vs Placebo (Randomized Treatment Period); Based on a Bayesian analysis of a sigmoidal dose-response relationship; Test type: Superiority; Odds Ratio (OR) = 1.422, 95% CI 2-sided [0.868 to 2.597]
Statistical Analysis 2: Comparison: FE 201836 350 ug (Randomized Treatment Period) vs Placebo (Randomized Treatment Period); Based on a Bayesian analysis of a sigmoidal dose-response relationship; Test type: Superiority; Odds Ratio (OR) = 1.373, 95% CI 2-sided [0.905 to 2.450]
Statistical Analysis 3: Comparison: FE 201836 250 ug (Randomized Treatment Period) vs Placebo (Randomized Treatment Period); Based on a Bayesian analysis of a sigmoidal dose-response relationship; Test type: Superiority; Odds Ratio (OR) = 1.284, 95% CI 2-sided [0.927 to 2.264]
Statistical Analysis 4: Comparison: FE 201836 150 ug (Randomized Treatment Period) vs Placebo (Randomized Treatment Period); Based on a Bayesian analysis of a sigmoidal dose-response relationship; Test type: Superiority; Odds Ratio (OR) = 1.145, 95% CI 2-sided [0.957 to 1.896]
Statistical Analysis 5: Comparison: FE 201836 100 ug (Randomized Treatment Period) vs Placebo (Randomized Treatment Period); Based on a Bayesian analysis of a sigmoidal dose-response relationship; Test type: Superiority; Odds Ratio (OR) = 1.079, 95% CI 2-sided [0.972 to 1.638]
Statistical Analysis 6: Comparison: FE 201836 50 ug (Randomized Treatment Period) vs Placebo (Randomized Treatment Period); Based on a Bayesian analysis of a sigmoidal dose-response relationship; Test type: Superiority; Odds Ratio (OR) = 1.023, 95% CI 2-sided [0.991 to 1.313]

11. Secondary Outcome: Change From Baseline in Mean NI Diary Total Score at Week 1
Description: The NI Diary is a 12-item questionnaire with 11 core items (Q1-Q11) and an overall quality of life (QoL) impact question (Q12). The NI Diary Total Scores are calculated by summing the 11 core items.Responses are scored from 0 to 4 (lowest t o highest impact). The NI Diary Total is standardized from 0 to 100 (lowest to highest impact).
  The score at each visit was calculated as the average over the three consecutive 24 hour periods just prior to the respective visit. Adjusted visit-specific mean changes from baseline in NI Diary Total Score are estimated using a baseline value of 40.
Time Frame: Baseline, Week 1
Population: The ITT-RT comprised of all the subjects randomized at Visit 4.
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | FE 201836 500 ug (Randomized Treatment Period) | FE 201836 350 ug (Randomized Treatment Period) | FE 201836 250 ug (Randomized Treatment Period) | FE 201836 150 ug (Randomized Treatment Period) | FE 201836 100 ug (Randomized Treatment Period) | FE 201836 50 ug (Randomized Treatment Period) | Placebo (Randomized Treatment Period)
Number analyzed (Participants) | 55 | 23 | 24 | 14 | 12 | 31 | 83
score on a scale | -7.55 [-11.67 to -3.43] | -21.91 [-28.15 to -15.68] | -10.90 [-17.17 to -4.63] | -8.93 [-17.15 to -0.72] | -9.68 [-18.41 to -0.94] | -8.75 [-14.27 to -3.23] | -8.07 [-11.48 to -4.65]
Statistical Analysis 1: Comparison: FE 201836 500 ug (Randomized Treatment Period) vs Placebo (Randomized Treatment Period); Test type: Superiority; p = 0.8463, MMRM — Threshold for significance at 0.05 level; Mean Difference = 0.52, 95% CI 2-sided [-4.75 to 5.78]
Statistical Analysis 2: Comparison: FE 201836 350 ug (Randomized Treatment Period) vs Placebo (Randomized Treatment Period); Test type: Superiority; p = 0.0001, MMRM — Threshold for significance at 0.05 level; Mean Difference = -13.85, 95% CI 2-sided [-20.89 to -6.81]
Statistical Analysis 3: Comparison: FE 201836 250 ug (Randomized Treatment Period) vs Placebo (Randomized Treatment Period); Test type: Superiority; p = 0.4355, MMRM — Threshold for significance at 0.05 level; Mean Difference = -2.84, 95% CI 2-sided [-9.99 to 4.32]
Statistical Analysis 4: Comparison: FE 201836 150 ug (Randomized Treatment Period) vs Placebo (Randomized Treatment Period); Test type: Superiority; p = 0.8483, MMRM — Threshold for significance at 0.05 level; Mean Difference = -0.87, 95% CI 2-sided [-9.79 to 8.06]
Statistical Analysis 5: Comparison: FE 201836 100 ug (Randomized Treatment Period) vs Placebo (Randomized Treatment Period); Test type: Superiority; p = 0.7336, MMRM — Threshold for significance at 0.05 level; Mean Difference = -1.61, 95% CI 2-sided [-10.91 to 7.69]
Statistical Analysis 6: Comparison: FE 201836 50 ug (Randomized Treatment Period) vs Placebo (Randomized Treatment Period); Test type: Superiority; p = 0.8347, MMRM — Threshold for significance at 0.05 level; Mean Difference = -0.69, 95% CI 2-sided [-7.15 to 5.78]

12. Secondary Outcome: Change From Baseline in Mean NI Diary Total Score at Week 4
Description: The NI Diary is a 12-item questionnaire with 11 core items (Q1-Q11) and an overall QoL impact question (Q12). The NI Diary Total Scores are calculated by summing the 11 core items. Responses are scored from 0 to 4 (lowest to highest impact). The NI Diary Total is standardized from 0 to 100 (lowest to highest impact).
  The score at each visit was calculated as the average over the three consecutive 24 hour periods just prior to the respective visit. Adjusted visit-specific mean changes from baseline in NI Diary Total Score are estimated using a baseline value of 40.
Time Frame: Baseline, Week 4
Population: The ITT-RT comprised of all the subjects randomized at Visit 4.
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | FE 201836 500 ug (Randomized Treatment Period) | FE 201836 350 ug (Randomized Treatment Period) | FE 201836 250 ug (Randomized Treatment Period) | FE 201836 150 ug (Randomized Treatment Period) | FE 201836 100 ug (Randomized Treatment Period) | FE 201836 50 ug (Randomized Treatment Period) | Placebo (Randomized Treatment Period)
Number analyzed (Participants) | 53 | 24 | 22 | 13 | 13 | 31 | 78
score on a scale | -12.62 [-16.89 to -8.35] | -17.44 [-23.80 to -11.08] | -14.37 [-20.96 to -7.78] | -11.23 [-19.82 to -2.65] | -22.23 [-31.11 to -13.35] | -13.29 [-19.00 to -7.58] | -14.20 [-17.77 to -10.64]
Statistical Analysis 1: Comparison: FE 201836 500 ug (Randomized Treatment Period) vs Placebo (Randomized Treatment Period); Test type: Superiority; p = 0.5695, MMRM — Threshold for significance at 0.05 level; Mean Difference = 1.59, 95% CI 2-sided [-3.90 to 7.07]
Statistical Analysis 2: Comparison: FE 201836 350 ug (Randomized Treatment Period) vs Placebo (Randomized Treatment Period); Test type: Superiority; p = 0.3784, MMRM — Threshold for significance at 0.05 level; Mean Difference = -3.23, 95% CI 2-sided [-10.46 to 3.99]
Statistical Analysis 3: Comparison: FE 201836 250 ug (Randomized Treatment Period) vs Placebo (Randomized Treatment Period); Test type: Superiority; p = 0.9653, MMRM — Threshold for significance at 0.05 level; Mean Difference = -0.17, 95% CI 2-sided [-7.67 to 7.34]
Statistical Analysis 4: Comparison: FE 201836 150 ug (Randomized Treatment Period) vs Placebo (Randomized Treatment Period); Test type: Superiority; p = 0.5304, MMRM — Threshold for significance at 0.05 level; Mean Difference = 2.97, 95% CI 2-sided [-6.35 to 12.29]
Statistical Analysis 5: Comparison: FE 201836 100 ug (Randomized Treatment Period) vs Placebo (Randomized Treatment Period); Test type: Superiority; p = 0.0968, MMRM — Threshold for significance at 0.05 level; Mean Difference = -8.02, 95% CI 2-sided [-17.51 to 1.46]
Statistical Analysis 6: Comparison: FE 201836 50 ug (Randomized Treatment Period) vs Placebo (Randomized Treatment Period); Test type: Superiority; p = 0.7885, MMRM — Threshold for significance at 0.05 level; Mean Difference = 0.91, 95% CI 2-sided [-5.79 to 7.62]

13. Secondary Outcome: Change From Baseline in Mean NI Diary Total Score at Week 8
Description: as for outcome 12
Time Frame: Baseline, Week 8
Population: The ITT-RT comprised of all the subjects randomized at Visit 4.
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | FE 201836 500 ug (Randomized Treatment Period) | FE 201836 350 ug (Randomized Treatment Period) | FE 201836 250 ug (Randomized Treatment Period) | FE 201836 150 ug (Randomized Treatment Period) | FE 201836 100 ug (Randomized Treatment Period) | FE 201836 50 ug (Randomized Treatment Period) | Placebo (Randomized Treatment Period)
Number analyzed (Participants) | 50 | 24 | 23 | 14 | 11 | 30 | 79
score on a scale | -16.03 [-20.49 to -11.57] | -23.22 [-29.79 to -16.64] | -15.10 [-21.85 to -8.35] | -12.04 [-20.77 to -3.32] | -19.23 [-28.62 to -9.83] | -14.11 [-20.00 to -8.22] | -14.83 [-18.50 to -11.16]
Statistical Analysis 1: Comparison: FE 201836 500 ug (Randomized Treatment Period) vs Placebo (Randomized Treatment Period); Test type: Superiority; p = 0.6792, MMRM — Threshold for significance at 0.05 level; Mean Difference = -1.20, 95% CI 2-sided [-6.89 to 4.50]
Statistical Analysis 2: Comparison: FE 201836 350 ug (Randomized Treatment Period) vs Placebo (Randomized Treatment Period); Test type: Superiority; p = 0.0276, MMRM — Threshold for significance at 0.05 level; Mean Difference = -8.39, 95% CI 2-sided [-15.84 to -0.93]
Statistical Analysis 3: Comparison: FE 201836 250 ug (Randomized Treatment Period) vs Placebo (Randomized Treatment Period); Test type: Superiority; p = 0.9445, MMRM — Threshold for significance at 0.05 level; Mean Difference = -0.27, 95% CI 2-sided [-7.97 to 7.42]
Statistical Analysis 4: Comparison: FE 201836 150 ug (Randomized Treatment Period) vs Placebo (Randomized Treatment Period); Test type: Superiority; p = 0.5637, MMRM — Threshold for significance at 0.05 level; Mean Difference = 2.79, 95% CI 2-sided [-6.71 to 12.28]
Statistical Analysis 5: Comparison: FE 201836 100 ug (Randomized Treatment Period) vs Placebo (Randomized Treatment Period); Test type: Superiority; p = 0.3870, MMRM — Threshold for significance at 0.05 level; Mean Difference = -4.40, 95% CI 2-sided [-14.39 to 5.60]
Statistical Analysis 6: Comparison: FE 201836 50 ug (Randomized Treatment Period) vs Placebo (Randomized Treatment Period); Test type: Superiority; p = 0.8373, MMRM — Threshold for significance at 0.05 level; Mean Difference = 0.72, 95% CI 2-sided [-6.19 to 7.63]

14. Secondary Outcome: Change From Baseline in Mean NI Diary Total Score at Week 12
Description: as for outcome 12
Time Frame: Baseline, Week 12
Population: The ITT-RT comprised of all the subjects randomized at Visit 4.
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | FE 201836 500 ug (Randomized Treatment Period) | FE 201836 350 ug (Randomized Treatment Period) | FE 201836 250 ug (Randomized Treatment Period) | FE 201836 150 ug (Randomized Treatment Period) | FE 201836 100 ug (Randomized Treatment Period) | FE 201836 50 ug (Randomized Treatment Period) | Placebo (Randomized Treatment Period)
Number analyzed (Participants) | 50 | 22 | 21 | 14 | 12 | 31 | 77
score on a scale | -16.92 [-21.66 to -12.18] | -24.44 [-31.52 to -17.35] | -14.68 [-21.94 to -7.42] | -10.13 [-19.37 to -0.88] | -22.59 [-32.46 to -12.71] | -17.18 [-23.39 to -10.96] | -17.45 [-21.36 to -13.53]
Statistical Analysis 1: Comparison: FE 201836 500 ug (Randomized Treatment Period) vs Placebo (Randomized Treatment Period); Test type: Superiority; p = 0.8646, MMRM — Threshold for significance at 0.05 level; Mean Difference = 0.53, 95% CI 2-sided [-5.54 to 6.59]
Statistical Analysis 2: Comparison: FE 201836 350 ug (Randomized Treatment Period) vs Placebo (Randomized Treatment Period); Test type: Superiority; p = 0.0870, MMRM — Threshold for significance at 0.05 level; Mean Difference = -6.99, 95% CI 2-sided [-15.00 to 1.02]
Statistical Analysis 3: Comparison: FE 201836 250 ug (Randomized Treatment Period) vs Placebo (Randomized Treatment Period); Test type: Superiority; p = 0.5100, MMRM — Threshold for significance at 0.05 level; Mean Difference = 2.77, 95% CI 2-sided [-5.50 to 11.04]
Statistical Analysis 4: Comparison: FE 201836 150 ug (Randomized Treatment Period) vs Placebo (Randomized Treatment Period); Test type: Superiority; p = 0.1535, MMRM — Threshold for significance at 0.05 level; Mean Difference = 7.32, 95% CI 2-sided [-2.75 to 17.39]
Statistical Analysis 5: Comparison: FE 201836 100 ug (Randomized Treatment Period) vs Placebo (Randomized Treatment Period); Test type: Superiority; p = 0.3369, MMRM — Threshold for significance at 0.05 level; Mean Difference = -5.14, 95% CI 2-sided [-15.66 to 5.38]
Statistical Analysis 6: Comparison: FE 201836 50 ug (Randomized Treatment Period) vs Placebo (Randomized Treatment Period); Test type: Superiority; p = 0.9417, MMRM — Threshold for significance at 0.05 level; Mean Difference = 0.27, 95% CI 2-sided [-7.05 to 7.59]

15. Secondary Outcome: Change From Baseline in Aggregated Mean NI Diary Total Score During 12 Weeks of Treatment
Description: The NI Diary is a 12-item questionnaire with 11 core items (Q1-Q11) and an overall QoL impact question (Q12). The NI Diary Total Scores are calculated by summing the 11 core items. Responses are scored from 0 to 4 (lowest to highest impact). The NI Diary Total is standardized from 0 to 100 (lowest to highest impact).
  The score at each visit was calculated as the mean over the three consecutive 24 hour periods just prior to the respective visit. The visit-specific means were aggregated into a mean of current and preceding visits.
  Level estimated for baseline value of mean NI Diary Total Score equal to 40 is presented in this endpoint.
  The 95% credibility interval (2.5 and 97.5 percentiles of the posterior distribution) instead of confidence interval is presented for this endpoint.
Time Frame: Baseline, during 12 weeks of treatment
Population: The ITT-RT comprised of all the subjects randomized at Visit 4.
Measure: Median (95% Confidence Interval); unit: score on a scale
Arm/Group | FE 201836 500 ug (Randomized Treatment Period) | FE 201836 350 ug (Randomized Treatment Period) | FE 201836 250 ug (Randomized Treatment Period) | FE 201836 150 ug (Randomized Treatment Period) | FE 201836 100 ug (Randomized Treatment Period) | FE 201836 50 ug (Randomized Treatment Period) | Placebo (Randomized Treatment Period)
Number analyzed (Participants) | 60 | 27 | 24 | 14 | 13 | 34 | 87
score on a scale | -12.40 [-14.71 to -8.59] | -12.69 [-15.07 to -10.53] | -12.75 [-15.16 to -10.57] | -12.77 [-15.21 to -10.59] | -12.77 [-15.23 to -10.54] | -12.78 [-15.18 to -10.50] | -12.77 [-15.18 to -10.47]
Statistical Analysis 1: Comparison: FE 201836 500 ug (Randomized Treatment Period) vs Placebo (Randomized Treatment Period); Based on a Bayesian analysis of a sigmoidal dose-response relationship; Test type: Superiority; Median difference = 0.00, 95% CI 2-sided [-1.41 to 5.47]
Statistical Analysis 2: Comparison: FE 201836 350 ug (Randomized Treatment Period) vs Placebo (Randomized Treatment Period); Based on a Bayesian analysis of a sigmoidal dose-response relationship; Test type: Superiority; Median difference = 0.00, 95% CI 2-sided [-0.43 to 1.19]
Statistical Analysis 3: Comparison: FE 201836 250 ug (Randomized Treatment Period) vs Placebo (Randomized Treatment Period); Based on a Bayesian analysis of a sigmoidal dose-response relationship; Test type: Superiority; Median difference = 0.00, 95% CI 2-sided [-0.16 to 0.50]
Statistical Analysis 4: Comparison: FE 201836 150 ug (Randomized Treatment Period) vs Placebo (Randomized Treatment Period); Based on a Bayesian analysis of a sigmoidal dose-response relationship; Test type: Superiority; Median difference = 0.00, 95% CI 2-sided [-0.03 to 0.15]
Statistical Analysis 5: Comparison: FE 201836 100 ug (Randomized Treatment Period) vs Placebo (Randomized Treatment Period); Based on a Bayesian analysis of a sigmoidal dose-response relationship; Test type: Superiority; Median difference = 0.00, 95% CI 2-sided [-0.01 to 0.05]
Statistical Analysis 6: Comparison: FE 201836 50 ug (Randomized Treatment Period) vs Placebo (Randomized Treatment Period); Based on a Bayesian analysis of a sigmoidal dose-response relationship; Test type: Superiority; Median difference = 0.00, 95% CI 2-sided [-0.00 to 0.01]

16. Secondary Outcome: Percentage of Nights With at Most One Nocturnal Void During 12 Weeks of Treatment
Description: The percentages of nights during the treatment period with at most one nocturnal void are presented in this endpoint.
  Level estimated for baseline value of mean number of nocturnal voids equal to 2 is presented in this endpoint.
Time Frame: During 12 weeks of treatment
Population: The ITT-RT comprised of all the subjects randomized at Visit 4.
Measure: Mean (95% Confidence Interval); unit: percentage of nights
Arm/Group | FE 201836 500 ug (Randomized Treatment Period) | FE 201836 350 ug (Randomized Treatment Period) | FE 201836 250 ug (Randomized Treatment Period) | FE 201836 150 ug (Randomized Treatment Period) | FE 201836 100 ug (Randomized Treatment Period) | FE 201836 50 ug (Randomized Treatment Period) | Placebo (Randomized Treatment Period)
Number analyzed (Participants) | 58 | 27 | 24 | 14 | 13 | 33 | 84
percentage of nights | 67.2 [58.2 to 76.2] | 77.5 [64.9 to 90.2] | 64.5 [51.0 to 78.0] | 55.3 [38.3 to 72.3] | 73.2 [55.1 to 91.2] | 61.4 [49.3 to 73.5] | 62.0 [53.8 to 70.2]
Statistical Analysis 1: Comparison: FE 201836 500 ug (Randomized Treatment Period) vs Placebo (Randomized Treatment Period); Test type: Superiority; p = 0.3328, ANCOVA — Threshold for significance at 0.05 level; Mean Difference = 5.2, 95% CI 2-sided [-5.3 to 15.7]
Statistical Analysis 2: Comparison: FE 201836 350 ug (Randomized Treatment Period) vs Placebo (Randomized Treatment Period); Test type: Superiority; p = 0.0255, ANCOVA — Threshold for significance at 0.05 level; Mean Difference = 15.5, 95% CI 2-sided [1.9 to 29.2]
Statistical Analysis 3: Comparison: FE 201836 250 ug (Randomized Treatment Period) vs Placebo (Randomized Treatment Period); Test type: Superiority; p = 0.7296, ANCOVA — Threshold for significance at 0.05 level; Mean Difference = 2.5, 95% CI 2-sided [-11.7 to 16.7]
Statistical Analysis 4: Comparison: FE 201836 150 ug (Randomized Treatment Period) vs Placebo (Randomized Treatment Period); Test type: Superiority; p = 0.4586, ANCOVA — Threshold for significance at 0.05 level; Mean Difference = -6.7, 95% CI 2-sided [-24.5 to 11.1]
Statistical Analysis 5: Comparison: FE 201836 100 ug (Randomized Treatment Period) vs Placebo (Randomized Treatment Period); Test type: Superiority; p = 0.2327, ANCOVA — Threshold for significance at 0.05 level; Mean Difference = 11.2, 95% CI 2-sided [-7.2 to 29.5]
Statistical Analysis 6: Comparison: FE 201836 50 ug (Randomized Treatment Period) vs Placebo (Randomized Treatment Period); Test type: Superiority; p = 0.9240, ANCOVA — Threshold for significance at 0.05 level; Mean Difference = -0.6, 95% CI 2-sided [-13.3 to 12.1]

17. Secondary Outcome: Percentage of Nights With No Nocturnal Voids During 12 Weeks of Treatment
Description: The percentages of nights during the treatment period with complete response, i.e. no nocturnal voids are presented in this endpoint.
  Level estimated for baseline value of mean number of nocturnal voids equal to 2 is presented in this endpoint.
Time Frame: During 12 weeks of treatment
Population: The ITT-RT comprised of all the subjects randomized at Visit 4.
Measure: Mean (95% Confidence Interval); unit: percentage of nights
Arm/Group | FE 201836 500 ug (Randomized Treatment Period) | FE 201836 350 ug (Randomized Treatment Period) | FE 201836 250 ug (Randomized Treatment Period) | FE 201836 150 ug (Randomized Treatment Period) | FE 201836 100 ug (Randomized Treatment Period) | FE 201836 50 ug (Randomized Treatment Period) | Placebo (Randomized Treatment Period)
Number analyzed (Participants) | 58 | 27 | 24 | 14 | 13 | 33 | 84
percentage of nights | 23.3 [16.3 to 30.3] | 28.8 [19.0 to 38.6] | 17.3 [6.8 to 27.8] | 12.9 [-0.3 to 26.1] | 14.8 [0.8 to 28.8] | 21.5 [12.1 to 30.9] | 23.0 [16.6 to 29.4]
Statistical Analysis 1: Comparison: FE 201836 500 ug (Randomized Treatment Period) vs Placebo (Randomized Treatment Period); Test type: Superiority; p = 0.9499, ANCOVA — Threshold for significance at 0.05 level; Mean Difference = 0.3, 95% CI 2-sided [-7.9 to 8.5]
Statistical Analysis 2: Comparison: FE 201836 350 ug (Randomized Treatment Period) vs Placebo (Randomized Treatment Period); Test type: Superiority; p = 0.2842, ANCOVA — Threshold for significance at 0.05 level; Mean Difference = 5.8, 95% CI 2-sided [-4.8 to 16.4]
Statistical Analysis 3: Comparison: FE 201836 250 ug (Randomized Treatment Period) vs Placebo (Randomized Treatment Period); Test type: Superiority; p = 0.3100, ANCOVA — Threshold for significance at 0.05 level; Mean Difference = -5.7, 95% CI 2-sided [-16.8 to 5.4]
Statistical Analysis 4: Comparison: FE 201836 150 ug (Randomized Treatment Period) vs Placebo (Randomized Treatment Period); Test type: Superiority; p = 0.1499, ANCOVA — Threshold for significance at 0.05 level; Mean Difference = -10.1, 95% CI 2-sided [-23.9 to 3.7]
Statistical Analysis 5: Comparison: FE 201836 100 ug (Randomized Treatment Period) vs Placebo (Randomized Treatment Period); Test type: Superiority; p = 0.2571, ANCOVA — Threshold for significance at 0.05 level; Mean Difference = -8.2, 95% CI 2-sided [-22.5 to 6.0]
Statistical Analysis 6: Comparison: FE 201836 50 ug (Randomized Treatment Period) vs Placebo (Randomized Treatment Period); Test type: Superiority; p = 0.7629, ANCOVA — Threshold for significance at 0.05 level; Mean Difference = -1.5, 95% CI 2-sided [-11.4 to 8.3]

18. Secondary Outcome: Change From Baseline in Mean NI Diary Overall Impact Score at Week 1
Description: The NI Diary is a 12-item questionnaire with 11 core items (Q1-Q11) and an overall QoL impact question (Q12). For the overall impact question (Q12), response options range from 0 (not at all) to 4 (a great deal). The NI Diary Overall Impact Scores are standardized from 0 to 100 (lowest to highest impact).
  The score at each visit was calculated as the average over the three consecutive 24 hour periods just prior to the respective visit. Adjusted visit-specific mean changes from baseline in NI Diary Overall Impact Score are estimated using a baseline value of 40.
Time Frame: Baseline, Week 1
Population: The ITT-RT comprised of all the subjects randomized at Visit 4.
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | FE 201836 500 ug (Randomized Treatment Period) | FE 201836 350 ug (Randomized Treatment Period) | FE 201836 250 ug (Randomized Treatment Period) | FE 201836 150 ug (Randomized Treatment Period) | FE 201836 100 ug (Randomized Treatment Period) | FE 201836 50 ug (Randomized Treatment Period) | Placebo (Randomized Treatment Period)
Number analyzed (Participants) | 55 | 23 | 24 | 14 | 12 | 31 | 83
score on a scale | -10.98 [-16.40 to -5.56] | -30.39 [-38.62 to -22.17] | -15.51 [-23.85 to -7.17] | -11.77 [-22.69 to -0.85] | -2.79 [-14.29 to 8.70] | -12.26 [-19.57 to -4.95] | -13.46 [-17.89 to -9.03]
Statistical Analysis 1: Comparison: FE 201836 500 ug (Randomized Treatment Period) vs Placebo (Randomized Treatment Period); Test type: Superiority; p = 0.4846, MMRM — Threshold for significance at 0.05 level; Mean Difference = 2.48, 95% CI 2-sided [-4.50 to 9.46]
Statistical Analysis 2: Comparison: FE 201836 350 ug (Randomized Treatment Period) vs Placebo (Randomized Treatment Period); Test type: Superiority; p = 0.0004, MMRM — Threshold for significance at 0.05 level; Mean Difference = -16.93, 95% CI 2-sided [-26.26 to -7.60]
Statistical Analysis 3: Comparison: FE 201836 250 ug (Randomized Treatment Period) vs Placebo (Randomized Treatment Period); Test type: Superiority; p = 0.6685, MMRM — Threshold for significance at 0.05 level; Mean Difference = -2.05, 95% CI 2-sided [-11.47 to 7.37]
Statistical Analysis 4: Comparison: FE 201836 150 ug (Randomized Treatment Period) vs Placebo (Randomized Treatment Period); Test type: Superiority; p = 0.7772, MMRM — Threshold for significance at 0.05 level; Mean Difference = 1.69, 95% CI 2-sided [-10.07 to 13.46]
Statistical Analysis 5: Comparison: FE 201836 100 ug (Randomized Treatment Period) vs Placebo (Randomized Treatment Period); Test type: Superiority; p = 0.0895, MMRM — Threshold for significance at 0.05 level; Mean Difference = 10.67, 95% CI 2-sided [-1.66 to 23.00]
Statistical Analysis 6: Comparison: FE 201836 50 ug (Randomized Treatment Period) vs Placebo (Randomized Treatment Period); Test type: Superiority; p = 0.7820, MMRM; Mean Difference = 1.20, 95% CI 2-sided [-7.34 to 9.74]

19. Secondary Outcome: Change From Baseline in Mean NI Diary Overall Impact Score at Week 4
Description: as for outcome 18
Time Frame: Baseline, Week 4
Population: The ITT-RT comprised of all the subjects randomized at Visit 4.
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | FE 201836 500 ug (Randomized Treatment Period) | FE 201836 350 ug (Randomized Treatment Period) | FE 201836 250 ug (Randomized Treatment Period) | FE 201836 150 ug (Randomized Treatment Period) | FE 201836 100 ug (Randomized Treatment Period) | FE 201836 50 ug (Randomized Treatment Period) | Placebo (Randomized Treatment Period)
Number analyzed (Participants) | 53 | 24 | 22 | 13 | 13 | 31 | 78
score on a scale | -22.17 [-28.25 to -16.09] | -26.07 [-35.09 to -17.05] | -19.35 [-28.80 to -9.90] | -18.36 [-30.66 to -6.07] | -17.95 [-30.50 to -5.41] | -21.40 [-29.54 to -13.26] | -21.75 [-26.74 to -16.77]
Statistical Analysis 1: Comparison: FE 201836 500 ug (Randomized Treatment Period) vs Placebo (Randomized Treatment Period); Test type: Superiority; p = 0.9175, MMRM — Threshold for significance at 0.05 level; Mean Difference = -0.41, 95% CI 2-sided [-8.25 to 7.42]
Statistical Analysis 2: Comparison: FE 201836 350 ug (Randomized Treatment Period) vs Placebo (Randomized Treatment Period); Test type: Superiority; p = 0.4098, MMRM — Threshold for significance at 0.05 level; Mean Difference = -4.32, 95% CI 2-sided [-14.62 to 5.98]
Statistical Analysis 3: Comparison: FE 201836 250 ug (Randomized Treatment Period) vs Placebo (Randomized Treatment Period); Test type: Superiority; p = 0.6566, MMRM — Threshold for significance at 0.05 level; Mean Difference = 2.41, 95% CI 2-sided [-8.25 to 13.06]
Statistical Analysis 4: Comparison: FE 201836 150 ug (Randomized Treatment Period) vs Placebo (Randomized Treatment Period); Test type: Superiority; p = 0.6144, MMRM — Threshold for significance at 0.05 level; Mean Difference = 3.39, 95% CI 2-sided [-9.85 to 16.63]
Statistical Analysis 5: Comparison: FE 201836 100 ug (Randomized Treatment Period) vs Placebo (Randomized Treatment Period); Test type: Superiority; p = 0.5798, MMRM — Threshold for significance at 0.05 level; Mean Difference = 3.80, 95% CI 2-sided [-9.71 to 17.31]
Statistical Analysis 6: Comparison: FE 201836 50 ug (Randomized Treatment Period) vs Placebo (Randomized Treatment Period); Test type: Superiority; p = 0.9417, MMRM — Threshold for significance at 0.05 level; Mean Difference = 0.35, 95% CI 2-sided [-9.17 to 9.88]

20. Secondary Outcome: Change From Baseline in Mean NI Diary Overall Impact Score at Week 8
Description: as for outcome 18
Time Frame: Baseline, Week 8
Population: The ITT-RT comprised of all the subjects randomized at Visit 4.
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | FE 201836 500 ug (Randomized Treatment Period) | FE 201836 350 ug (Randomized Treatment Period) | FE 201836 250 ug (Randomized Treatment Period) | FE 201836 150 ug (Randomized Treatment Period) | FE 201836 100 ug (Randomized Treatment Period) | FE 201836 50 ug (Randomized Treatment Period) | Placebo (Randomized Treatment Period)
Number analyzed (Participants) | 50 | 24 | 23 | 14 | 11 | 30 | 79
score on a scale | -28.13 [-34.76 to -21.50] | -34.97 [-44.69 to -25.25] | -21.71 [-31.80 to -11.62] | -19.03 [-32.06 to -6.00] | -23.84 [-37.71 to -9.96] | -20.70 [-29.45 to -11.94] | -25.32 [-30.69 to -19.95]
Statistical Analysis 1: Comparison: FE 201836 500 ug (Randomized Treatment Period) vs Placebo (Randomized Treatment Period); Test type: Superiority; p = 0.5148, MMRM — Threshold for significance at 0.05 level; Mean Difference = -2.81, 95% CI 2-sided [-11.31 to 5.68]
Statistical Analysis 2: Comparison: FE 201836 350 ug (Randomized Treatment Period) vs Placebo (Randomized Treatment Period); Test type: Superiority; p = 0.0879, MMRM — Threshold for significance at 0.05 level; Mean Difference = -9.65, 95% CI 2-sided [-20.75 to 1.44]
Statistical Analysis 3: Comparison: FE 201836 250 ug (Randomized Treatment Period) vs Placebo (Randomized Treatment Period); Test type: Superiority; p = 0.5335, MMRM — Threshold for significance at 0.05 level; Mean Difference = 3.61, 95% CI 2-sided [-7.79 to 15.00]
Statistical Analysis 4: Comparison: FE 201836 150 ug (Randomized Treatment Period) vs Placebo (Randomized Treatment Period); Test type: Superiority; p = 0.3787, MMRM — Threshold for significance at 0.05 level; Mean Difference = 6.29, 95% CI 2-sided [-7.76 to 20.34]
Statistical Analysis 5: Comparison: FE 201836 100 ug (Randomized Treatment Period) vs Placebo (Randomized Treatment Period); Test type: Superiority; p = 0.8448, MMRM — Threshold for significance at 0.05 level; Mean Difference = 1.48, 95% CI 2-sided [-13.41 to 16.38]
Statistical Analysis 6: Comparison: FE 201836 50 ug (Randomized Treatment Period) vs Placebo (Randomized Treatment Period); Test type: Superiority; p = 0.3751, MMRM — Threshold for significance at 0.05 level; Mean Difference = 4.62, 95% CI 2-sided [-5.63 to 14.87]

21. Secondary Outcome: Change From Baseline in Mean NI Diary Overall Impact Score at Week 12
Description: as for outcome 18
Time Frame: Baseline, Week 12
Population: The ITT-RT comprised of all the subjects randomized at Visit 4.
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | FE 201836 500 ug (Randomized Treatment Period) | FE 201836 350 ug (Randomized Treatment Period) | FE 201836 250 ug (Randomized Treatment Period) | FE 201836 150 ug (Randomized Treatment Period) | FE 201836 100 ug (Randomized Treatment Period) | FE 201836 50 ug (Randomized Treatment Period) | Placebo (Randomized Treatment Period)
Number analyzed (Participants) | 50 | 22 | 21 | 14 | 12 | 31 | 77
score on a scale | -30.47 [-37.49 to -23.45] | -36.76 [-47.18 to -26.34] | -20.84 [-31.65 to -10.02] | -15.32 [-29.10 to -1.54] | -28.89 [-43.40 to -14.39] | -27.13 [-36.35 to -17.91] | -30.03 [-35.74 to -24.33]
Statistical Analysis 1: Comparison: FE 201836 500 ug (Randomized Treatment Period) vs Placebo (Randomized Treatment Period); Test type: Superiority; p = 0.9245, MMRM — Threshold for significance at 0.05 level; Mean Difference = -0.43, 95% CI 2-sided [-9.43 to 8.57]
Statistical Analysis 2: Comparison: FE 201836 350 ug (Randomized Treatment Period) vs Placebo (Randomized Treatment Period); Test type: Superiority; p = 0.2657, MMRM — Threshold for significance at 0.05 level; Mean Difference = -6.72, 95% CI 2-sided [-18.59 to 5.15]
Statistical Analysis 3: Comparison: FE 201836 250 ug (Randomized Treatment Period) vs Placebo (Randomized Treatment Period); Test type: Superiority; p = 0.1383, MMRM — Threshold for significance at 0.05 level; Mean Difference = 9.20, 95% CI 2-sided [-2.99 to 21.38]
Statistical Analysis 4: Comparison: FE 201836 150 ug (Randomized Treatment Period) vs Placebo (Randomized Treatment Period); Test type: Superiority; p = 0.0523, MMRM — Threshold for significance at 0.05 level; Mean Difference = 14.72, 95% CI 2-sided [-0.15 to 29.59]
Statistical Analysis 5: Comparison: FE 201836 100 ug (Randomized Treatment Period) vs Placebo (Randomized Treatment Period); Test type: Superiority; p = 0.8855, MMRM — Threshold for significance at 0.05 level; Mean Difference = 1.14, 95% CI 2-sided [-14.47 to 16.75]
Statistical Analysis 6: Comparison: FE 201836 50 ug (Randomized Treatment Period) vs Placebo (Randomized Treatment Period); Test type: Superiority; p = 0.5972, MMRM — Threshold for significance at 0.05 level; Mean Difference = 2.91, 95% CI 2-sided [-7.91 to 13.72]

22. Secondary Outcome: Change From Baseline in Aggregated Mean NI Diary Overall Impact Score During 12 Weeks of Treatment
Description: The NI Diary is a 12-item questionnaire with 11 core items (Q1-Q11) and an overall QoL impact question (Q12). For the overall impact question (Q12), response options range from 0 (not at all) to 4 (a great deal). The NI Diary Overall Impact Scores are standardized from 0 to 100 (lowest to highest impact).
  The score at each visit was calculated as the average over the three consecutive 24 hour periods just prior to the respective visit. The visit-specific means were aggregated into a mean of current and preceding visits.
  Level estimated for baseline value of mean NI Diary Overall Impact Score equal to 40 is presented in this endpoint.
  The 95% credibility interval (2.5 and 97.5 percentiles of the posterior distribution) instead of confidence interval is presented for this endpoint.
Time Frame: Baseline, during 12 weeks of treatment
Population: The ITT-RT comprised of all the subjects randomized at Visit 4.
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | FE 201836 500 ug (Randomized Treatment Period) | FE 201836 350 ug (Randomized Treatment Period) | FE 201836 250 ug (Randomized Treatment Period) | FE 201836 150 ug (Randomized Treatment Period) | FE 201836 100 ug (Randomized Treatment Period) | FE 201836 50 ug (Randomized Treatment Period) | Placebo (Randomized Treatment Period)
Number analyzed (Participants) | 60 | 27 | 24 | 14 | 13 | 34 | 87
score on a scale | -6.50 [-10.57 to -2.85] | -6.25 [-9.78 to -3.03] | -6.11 [-9.49 to -2.90] | -6.00 [-9.28 to -2.70] | -5.98 [-9.29 to -2.58] | -5.97 [-9.32 to -2.57] | -5.96 [-9.42 to -2.49]
Statistical Analysis 1: Comparison: FE 201836 500 ug (Randomized Treatment Period) vs Placebo (Randomized Treatment Period); Based on a Bayesian analysis of a sigmoidal dose-response relationship; Test type: Superiority; Mean Difference = -0.54, 95% CI 2-sided [-6.09 to 2.28]
Statistical Analysis 2: Comparison: FE 201836 350 ug (Randomized Treatment Period) vs Placebo (Randomized Treatment Period); Based on a Bayesian analysis of a sigmoidal dose-response relationship; Test type: Superiority; Mean Difference = -0.28, 95% CI 2-sided [-4.30 to 0.75]
Statistical Analysis 3: Comparison: FE 201836 250 ug (Randomized Treatment Period) vs Placebo (Randomized Treatment Period); Based on a Bayesian analysis of a sigmoidal dose-response relationship; Test type: Superiority; Mean Difference = -0.15, 95% CI 2-sided [-2.44 to 0.33]
Statistical Analysis 4: Comparison: FE 201836 150 ug (Randomized Treatment Period) vs Placebo (Randomized Treatment Period); Based on a Bayesian analysis of a sigmoidal dose-response relationship; Test type: Superiority; Mean Difference = -0.04, 95% CI 2-sided [-0.92 to 0.07]
Statistical Analysis 5: Comparison: FE 201836 100 ug (Randomized Treatment Period) vs Placebo (Randomized Treatment Period); Based on a Bayesian analysis of a sigmoidal dose-response relationship; Test type: Superiority; Mean Difference = -0.02, 95% CI 2-sided [-0.48 to 0.02]
Statistical Analysis 6: Comparison: FE 201836 50 ug (Randomized Treatment Period) vs Placebo (Randomized Treatment Period); Based on a Bayesian analysis of a sigmoidal dose-response relationship; Test type: Superiority; Mean Difference = -0.00, 95% CI 2-sided [-0.15 to 0.00]

23. Secondary Outcome: Patient Global Impression of Improvement (PGI-I) Urinary Symptoms Scores at Week 1
Description: The PGI-I is a 1-item questionnaire designed to assess the patient's impression of changes in urinary symptoms. The PGI-I was scored from 1 (very much better) to 7 (very much worse).
  Visit-specific PGI-I in urinary symptoms is presented in this endpoint.
Time Frame: Week 1
Population: The ITT-RT comprised of all the subjects randomized at Visit 4.
Measure: Mean (95% Confidence Interval); unit: score on a scale
Groups:
- FE 201836 50 ug (Randomized Treatment Period): FE 201836 50 µg oral solution and placebo ODT, administered once dail
Arm/Group | FE 201836 500 ug (Randomized Treatment Period) | FE 201836 350 ug (Randomized Treatment Period) | FE 201836 250 ug (Randomized Treatment Period) | FE 201836 150 ug (Randomized Treatment Period) | FE 201836 100 ug (Randomized Treatment Period) | FE 201836 50 ug (Randomized Treatment Period) | Placebo (Randomized Treatment Period)
Number analyzed (Participants) | 53 | 23 | 24 | 14 | 11 | 33 | 81
score on a scale | 2.475 [2.261 to 2.689] | 2.045 [1.723 to 2.367] | 2.708 [2.385 to 3.031] | 2.786 [2.363 to 3.209] | 2.781 [2.316 to 3.245] | 2.758 [2.482 to 3.033] | 2.745 [2.571 to 2.919]
Statistical Analysis 1: Comparison: FE 201836 500 ug (Randomized Treatment Period) vs Placebo (Randomized Treatment Period); Test type: Superiority; p = 0.0550, MMRM — Threshold for significance at 0.05 level; Mean Difference = -0.270, 95% CI 2-sided [-0.545 to 0.006]
Statistical Analysis 2: Comparison: FE 201836 350 ug (Randomized Treatment Period) vs Placebo (Randomized Treatment Period); Test type: Superiority; p = 0.0002, MMRM — Threshold for significance at 0.05 level; Mean Difference = -0.700, 95% CI 2-sided [-1.066 to -0.335]
Statistical Analysis 3: Comparison: FE 201836 250 ug (Randomized Treatment Period) vs Placebo (Randomized Treatment Period); Test type: Superiority; p = 0.8440, MMRM — Threshold for significance at 0.05 level; Mean Difference = -0.037, 95% CI 2-sided [-0.404 to 0.330]
Statistical Analysis 4: Comparison: FE 201836 150 ug (Randomized Treatment Period) vs Placebo (Randomized Treatment Period); Test type: Superiority; p = 0.8610, MMRM — Threshold for significance at 0.05 level; Mean Difference = 0.041, 95% CI 2-sided [-0.417 to 0.498]
Statistical Analysis 5: Comparison: FE 201836 100 ug (Randomized Treatment Period) vs Placebo (Randomized Treatment Period); Test type: Superiority; p = 0.8871, MMRM — Threshold for significance at 0.05 level; Mean Difference = 0.036, 95% CI 2-sided [-0.460 to 0.532]
Statistical Analysis 6: Comparison: FE 201836 50 ug (Randomized Treatment Period) vs Placebo (Randomized Treatment Period); Test type: Superiority; p = 0.9396, MMRM — Threshold for significance at 0.05 level; Mean Difference = 0.013, 95% CI 2-sided [-0.313 to 0.338]

24. Secondary Outcome: Patient Global Impression of Improvement (PGI-I) Urinary Symptoms Scores at Week 4
Description: as for outcome 23
Time Frame: Week 4
Population: The ITT-RT comprised of all the subjects randomized at Visit 4.
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | FE 201836 500 ug (Randomized Treatment Period) | FE 201836 350 ug (Randomized Treatment Period) | FE 201836 250 ug (Randomized Treatment Period) | FE 201836 150 ug (Randomized Treatment Period) | FE 201836 100 ug (Randomized Treatment Period) | FE 201836 50 ug (Randomized Treatment Period) | Placebo (Randomized Treatment Period)
Number analyzed (Participants) | 53 | 24 | 20 | 12 | 13 | 30 | 77
score on a scale | 2.121 [1.866 to 2.376] | 2.191 [1.813 to 2.569] | 2.447 [2.039 to 2.855] | 2.521 [1.995 to 3.047] | 2.385 [1.859 to 2.910] | 2.582 [2.244 to 2.921] | 2.596 [2.386 to 2.806]
Statistical Analysis 1: Comparison: FE 201836 500 ug (Randomized Treatment Period) vs Placebo (Randomized Treatment Period); Test type: Superiority; p = 0.0050, MMRM — Threshold for significance at 0.05 level; Mean Difference = -0.475, 95% CI 2-sided [-0.806 to -0.145]
Statistical Analysis 2: Comparison: FE 201836 350 ug (Randomized Treatment Period) vs Placebo (Randomized Treatment Period); Test type: Superiority; p = 0.0665, MMRM — Threshold for significance at 0.05 level; Mean Difference = -0.405, 95% CI 2-sided [-0.837 to 0.028]
Statistical Analysis 3: Comparison: FE 201836 250 ug (Randomized Treatment Period) vs Placebo (Randomized Treatment Period); Test type: Superiority; p = 0.5245, MMRM — Threshold for significance at 0.05 level; Mean Difference = -0.149, 95% CI 2-sided [-0.608 to 0.310]
Statistical Analysis 4: Comparison: FE 201836 150 ug (Randomized Treatment Period) vs Placebo (Randomized Treatment Period); Test type: Superiority; p = 0.7947, MMRM — Threshold for significance at 0.05 level; Mean Difference = -0.075, 95% CI 2-sided [-0.642 to 0.492]
Statistical Analysis 5: Comparison: FE 201836 100 ug (Randomized Treatment Period) vs Placebo (Randomized Treatment Period); Test type: Superiority; p = 0.4625, MMRM — Threshold for significance at 0.05 level; Mean Difference = -0.211, 95% CI 2-sided [-0.777 to 0.355]
Statistical Analysis 6: Comparison: FE 201836 50 ug (Randomized Treatment Period) vs Placebo (Randomized Treatment Period); Test type: Superiority; p = 0.9465, MMRM — Threshold for significance at 0.05 level; Mean Difference = -0.014, 95% CI 2-sided [-0.412 to 0.385]

25. Secondary Outcome: Patient Global Impression of Improvement (PGI-I) Urinary Symptoms Scores at Week 8
Description: as for outcome 23
Time Frame: Week 8
Population: The ITT-RT comprised of all the subjects randomized at Visit 4.
Measure: Mean (95% Confidence Interval); unit: score on a scale
Groups:
- FE 201836 350 ug (Randomized Treatment Period): FE 201836 500 µg oral solution and placebo ODT, administered once daily
Arm/Group | FE 201836 500 ug (Randomized Treatment Period) | FE 201836 350 ug (Randomized Treatment Period) | FE 201836 250 ug (Randomized Treatment Period) | FE 201836 150 ug (Randomized Treatment Period) | FE 201836 100 ug (Randomized Treatment Period) | FE 201836 50 ug (Randomized Treatment Period) | Placebo (Randomized Treatment Period)
Number analyzed (Participants) | 49 | 24 | 21 | 14 | 11 | 28 | 78
score on a scale | 1.843 [1.572 to 2.113] | 1.887 [1.493 to 2.281] | 2.528 [2.109 to 2.947] | 2.286 [1.761 to 2.811] | 2.155 [1.587 to 2.723] | 2.273 [1.917 to 2.629] | 2.573 [2.355 to 2.791]
Statistical Analysis 1: Comparison: FE 201836 500 ug (Randomized Treatment Period) vs Placebo (Randomized Treatment Period); Test type: Superiority; p < 0.0001, MMRM — Threshold for significance at 0.05 level; Mean Difference = -0.730, 95% CI 2-sided [-1.078 to -0.383]
Statistical Analysis 2: Comparison: FE 201836 350 ug (Randomized Treatment Period) vs Placebo (Randomized Treatment Period); Test type: Superiority; p = 0.0030, MMRM — Threshold for significance at 0.05 level; Mean Difference = -0.686, 95% CI 2-sided [-1.137 to -0.236]
Statistical Analysis 3: Comparison: FE 201836 250 ug (Randomized Treatment Period) vs Placebo (Randomized Treatment Period); Test type: Superiority; p = 0.8520, MMRM — Threshold for significance at 0.05 level; Mean Difference = -0.045, 95% CI 2-sided [-0.517 to 0.427]
Statistical Analysis 4: Comparison: FE 201836 150 ug (Randomized Treatment Period) vs Placebo (Randomized Treatment Period); Test type: Superiority; p = 0.3205, MMRM — Threshold for significance at 0.05 level; Mean Difference = -0.287, 95% CI 2-sided [-0.856 to 0.281]
Statistical Analysis 5: Comparison: FE 201836 100 ug (Randomized Treatment Period) vs Placebo (Randomized Treatment Period); Test type: Superiority; p = 0.1769, MMRM — Threshold for significance at 0.05 level; Mean Difference = -0.418, 95% CI 2-sided [-1.026 to 0.190]
Statistical Analysis 6: Comparison: FE 201836 50 ug (Randomized Treatment Period) vs Placebo (Randomized Treatment Period); Test type: Superiority; p = 0.1584, MMRM — Threshold for significance at 0.05 level; Mean Difference = -0.300, 95% CI 2-sided [-0.717 to 0.118]

26. Secondary Outcome: Patient Global Impression of Improvement (PGI-I) Urinary Symptoms Scores at Week 12
Description: as for outcome 23
Time Frame: Week 12
Population: The ITT-RT comprised of all the subjects randomized at Visit 4.
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | FE 201836 500 ug (Randomized Treatment Period) | FE 201836 350 ug (Randomized Treatment Period) | FE 201836 250 ug (Randomized Treatment Period) | FE 201836 150 ug (Randomized Treatment Period) | FE 201836 100 ug (Randomized Treatment Period) | FE 201836 50 ug (Randomized Treatment Period) | Placebo (Randomized Treatment Period)
Number analyzed (Participants) | 46 | 23 | 18 | 13 | 12 | 31 | 72
score on a scale | 1.667 [1.357 to 1.977] | 1.671 [1.224 to 2.119] | 2.656 [2.167 to 3.146] | 2.452 [1.855 to 3.049] | 1.678 [1.052 to 2.304] | 2.384 [1.994 to 2.774] | 2.490 [2.240 to 2.740]
Statistical Analysis 1: Comparison: FE 201836 500 ug (Randomized Treatment Period) vs Placebo (Randomized Treatment Period); Test type: Superiority; p < 0.0001, MMRM — Threshold for significance at 0.05 level; Mean Difference = -0.822, 95% CI 2-sided [-1.220 to -0.424]
Statistical Analysis 2: Comparison: FE 201836 350 ug (Randomized Treatment Period) vs Placebo (Randomized Treatment Period); Test type: Superiority; p = 0.0019, MMRM — Threshold for significance at 0.05 level; Mean Difference = -0.818, 95% CI 2-sided [-1.331 to -0.306]
Statistical Analysis 3: Comparison: FE 201836 250 ug (Randomized Treatment Period) vs Placebo (Randomized Treatment Period); Test type: Superiority; p = 0.5510, MMRM — Threshold for significance at 0.05 level; Mean Difference = 0.167, 95% CI 2-sided [-0.383 to 0.716]
Statistical Analysis 4: Comparison: FE 201836 150 ug (Randomized Treatment Period) vs Placebo (Randomized Treatment Period); Test type: Superiority; p = 0.9086, MMRM — Threshold for significance at 0.05 level; Mean Difference = -0.038, 95% CI 2-sided [-0.685 to 0.610]
Statistical Analysis 5: Comparison: FE 201836 100 ug (Randomized Treatment Period) vs Placebo (Randomized Treatment Period); Test type: Superiority; p = 0.0185, MMRM — Threshold for significance at 0.05 level; Mean Difference = -0.812, 95% CI 2-sided [-1.486 to -0.138]
Statistical Analysis 6: Comparison: FE 201836 50 ug (Randomized Treatment Period) vs Placebo (Randomized Treatment Period); Test type: Superiority; p = 0.6537, MMRM — Threshold for significance at 0.05 level; Mean Difference = -0.106, 95% CI 2-sided [-0.569 to 0.357]

27. Secondary Outcome: Change From Baseline in Patient Global Impression of Severity (PGI-S) Scores at Week 1
Description: The PGI-S is a 1-item questionnaire designed to assess patient's impression of disease severity. The PGI-S was scored from 1 (none) to 4 (severe).
  Change from baseline in visit-specific PGI-S is presented in this endpoint.
  Level estimated for baseline value of PGI-S equal to 3 is presented in this endpoint.
Time Frame: Baseline, Week 1
Population: The ITT-RT comprised of all the subjects randomized at Visit 4.
Measure: Least Squares Mean (95% Confidence Interval); unit: score on a scale
Groups:
- FE 201836 500 ug (Randomized Treatment Period): FE 201836 500 μg oral solution and placebo ODT, administered once daily
- FE 201836 350 ug (Randomized Treatment Period): FE 201836 350 μg oral solution and placebo ODT, administered once daily
- FE 201836 250 ug (Randomized Treatment Period): FE 201836 250 μg oral solution and placebo ODT, administered once daily
- FE 201836 150 ug (Randomized Treatment Period): FE 201836 150 μg oral solution and placebo ODT, administered once daily
- FE 201836 100 ug (Randomized Treatment Period): FE 201836 100 μg oral solution and placebo ODT, administered once daily
- FE 201836 50 ug (Randomized Treatment Period): FE 201836 50 μg oral solution and placebo ODT, administered once daily
Arm/Group | FE 201836 500 ug (Randomized Treatment Period) | FE 201836 350 ug (Randomized Treatment Period) | FE 201836 250 ug (Randomized Treatment Period) | FE 201836 150 ug (Randomized Treatment Period) | FE 201836 100 ug (Randomized Treatment Period) | FE 201836 50 ug (Randomized Treatment Period) | Placebo (Randomized Treatment Period)
Number analyzed (Participants) | 53 | 23 | 24 | 14 | 10 | 28 | 80
score on a scale | -0.739 [-0.927 to -0.552] | -0.970 [-1.253 to -0.688] | -0.811 [-1.094 to -0.529] | -0.643 [-1.012 to -0.273] | -0.417 [-0.840 to 0.007] | -0.719 [-0.984 to -0.454] | -0.593 [-0.746 to -0.440]
Statistical Analysis 1: Comparison: FE 201836 500 ug (Randomized Treatment Period) vs Placebo (Randomized Treatment Period); Test type: Superiority; p = 0.2350, MMRM — Threshold for significance at 0.05 level; Least Square Mean Difference = -0.146, 95% CI 2-sided [-0.388 to 0.096]
Statistical Analysis 2: Comparison: FE 201836 350 ug (Randomized Treatment Period) vs Placebo (Randomized Treatment Period); Test type: Superiority; p = 0.0215, MMRM — Threshold for significance at 0.05 level; Least Square Mean Difference = -0.377, 95% CI 2-sided [-0.699 to -0.056]
Statistical Analysis 3: Comparison: FE 201836 250 ug (Randomized Treatment Period) vs Placebo (Randomized Treatment Period); Test type: Superiority; p = 0.1818, MMRM — Threshold for significance at 0.05 level; Least Square Mean Difference = -0.218, 95% CI 2-sided [-0.540 to 0.103]
Statistical Analysis 4: Comparison: FE 201836 150 ug (Randomized Treatment Period) vs Placebo (Randomized Treatment Period); Test type: Superiority; p = 0.8063, MMRM — Threshold for significance at 0.05 level; Least Square Mean Difference = -0.050, 95% CI 2-sided [-0.450 to 0.350]
Statistical Analysis 5: Comparison: FE 201836 100 ug (Randomized Treatment Period) vs Placebo (Randomized Treatment Period); Test type: Superiority; p = 0.4414, MMRM — Threshold for significance at 0.05 level; Least Square Mean Difference = 0.176, 95% CI 2-sided [-0.274 to 0.627]
Statistical Analysis 6: Comparison: FE 201836 50 ug (Randomized Treatment Period) vs Placebo (Randomized Treatment Period); Test type: Superiority; p = 0.4179, MMRM — Threshold for significance at 0.05 level; Least Square Mean Difference = -0.126, 95% CI 2-sided [-0.432 to 0.180]

28. Secondary Outcome: Change From Baseline in PGI-S Scores at Week 4
Description: as for outcome 27
Time Frame: Baseline, Week 4
Population: The ITT-RT comprised of all the subjects randomized at Visit 4.
Measure: Least Squares Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | FE 201836 500 ug (Randomized Treatment Period) | FE 201836 350 ug (Randomized Treatment Period) | FE 201836 250 ug (Randomized Treatment Period) | FE 201836 150 ug (Randomized Treatment Period) | FE 201836 100 ug (Randomized Treatment Period) | FE 201836 50 ug (Randomized Treatment Period) | Placebo (Randomized Treatment Period)
Number analyzed (Participants) | 52 | 23 | 20 | 12 | 12 | 27 | 75
score on a scale | -0.837 [-1.015 to -0.659] | -1.025 [-1.292 to -0.758] | -0.798 [-1.081 to -0.516] | -0.749 [-1.115 to -0.383] | -0.656 [-1.033 to -0.278] | -0.936 [-1.189 to -0.684] | -0.898 [-1.045 to -0.750]
Statistical Analysis 1: Comparison: FE 201836 500 ug (Randomized Treatment Period) vs Placebo (Randomized Treatment Period); Test type: Superiority; p = 0.6042, MMRM — Threshold for significance at 0.05 level; Least Square Mean Difference = 0.061, 95% CI 2-sided [-0.170 to 0.292]
Statistical Analysis 2: Comparison: FE 201836 350 ug (Randomized Treatment Period) vs Placebo (Randomized Treatment Period); Test type: Superiority; p = 0.4114, MMRM — Threshold for significance at 0.05 level; Least Square Mean Difference = -0.127, 95% CI 2-sided [-0.432 to 0.177]
Statistical Analysis 3: Comparison: FE 201836 250 ug (Randomized Treatment Period) vs Placebo (Randomized Treatment Period); Test type: Superiority; p = 0.5394, MMRM — Threshold for significance at 0.05 level; Least Square Mean Difference = 0.099, 95% CI 2-sided [-0.219 to 0.418]
Statistical Analysis 4: Comparison: FE 201836 150 ug (Randomized Treatment Period) vs Placebo (Randomized Treatment Period); Test type: Superiority; p = 0.4590, MMRM — Threshold for significance at 0.05 level; Least Square Mean Difference = 0.149, 95% CI 2-sided [-0.246 to 0.544]
Statistical Analysis 5: Comparison: FE 201836 100 ug (Randomized Treatment Period) vs Placebo (Randomized Treatment Period); Test type: Superiority; p = 0.2397, MMRM — Threshold for significance at 0.05 level; Least Square Mean Difference = 0.242, 95% CI 2-sided [-0.163 to 0.647]
Statistical Analysis 6: Comparison: FE 201836 50 ug (Randomized Treatment Period) vs Placebo (Randomized Treatment Period); Test type: Superiority; p = 0.7954, MMRM — Threshold for significance at 0.05 level; Least Square Mean Difference = -0.039, 95% CI 2-sided [-0.332 to 0.254]

29. Secondary Outcome: Change From Baseline in PGI-S Scores at Week 8
Description: as for outcome 27
Time Frame: Baseline, Week 8
Population: The ITT-RT comprised of all the subjects randomized at Visit 4.
Measure: Least Squares Mean (95% Confidence Interval); unit: score on a scale
Groups:
- FE 201836 500 ug (Randomized Treatment Period): FE 201836 500 µg oral solution for daily intake
- FE 201836 350 ug (Randomized Treatment Period): FE 201836 350 µg oral solution for daily intake
- FE 201836 250 ug (Randomized Treatment Period): FE 201836 250 µg oral solution for daily intake
- FE 201836 150 ug (Randomized Treatment Period): FE 201836 150 µg oral solution for daily intake
- FE 201836 100 ug (Randomized Treatment Period): FE 201836 100 µg oral solution for daily intake
- FE 201836 50 ug (Randomized Treatment Period): FE 201836 50 µg oral solution for daily intake
- Placebo (Randomized Treatment Period): Placebo ODT, mimics active comparator drug
Arm/Group | FE 201836 500 ug (Randomized Treatment Period) | FE 201836 350 ug (Randomized Treatment Period) | FE 201836 250 ug (Randomized Treatment Period) | FE 201836 150 ug (Randomized Treatment Period) | FE 201836 100 ug (Randomized Treatment Period) | FE 201836 50 ug (Randomized Treatment Period) | Placebo (Randomized Treatment Period)
Number analyzed (Participants) | 48 | 23 | 21 | 14 | 11 | 25 | 76
score on a scale | -1.132 [-1.322 to -0.942] | -1.410 [-1.688 to -1.132] | -0.825 [-1.114 to -0.536] | -0.643 [-1.004 to -0.281] | -0.816 [-1.215 to -0.418] | -1.013 [-1.279 to -0.747] | -0.800 [-0.953 to -0.647]
Statistical Analysis 1: Comparison: FE 201836 500 ug (Randomized Treatment Period) vs Placebo (Randomized Treatment Period); Test type: Superiority; p = 0.0077, MMRM — Threshold for significance at 0.05 level; Least Square Mean Difference = -0.332, 95% CI 2-sided [-0.576 to -0.089]
Statistical Analysis 2: Comparison: FE 201836 350 ug (Randomized Treatment Period) vs Placebo (Randomized Treatment Period); Test type: Superiority; p = 0.0002, MMRM — Threshold for significance at 0.05 level; Least Square Mean Difference = -0.610, 95% CI 2-sided [-0.927 to -0.293]
Statistical Analysis 3: Comparison: FE 201836 250 ug (Randomized Treatment Period) vs Placebo (Randomized Treatment Period); Test type: Superiority; p = 0.8778, MMRM — Threshold for significance at 0.05 level; Least Square Mean Difference = -0.026, 95% CI 2-sided [-0.352 to 0.301]
Statistical Analysis 4: Comparison: FE 201836 150 ug (Randomized Treatment Period) vs Placebo (Randomized Treatment Period); Test type: Superiority; p = 0.4309, MMRM — Threshold for significance at 0.05 level; Least Square Mean Difference = 0.157, 95% CI 2-sided [-0.235 to 0.549]
Statistical Analysis 5: Comparison: FE 201836 100 ug (Randomized Treatment Period) vs Placebo (Randomized Treatment Period); Test type: Superiority; p = 0.9392, MMRM — Threshold for significance at 0.05 level; Least Square Mean Difference = -0.017, 95% CI 2-sided [-0.444 to 0.411]
Statistical Analysis 6: Comparison: FE 201836 50 ug (Randomized Treatment Period) vs Placebo (Randomized Treatment Period); Test type: Superiority; p = 0.1734, MMRM — Threshold for significance at 0.05 level; Least Square Mean Difference = -0.213, 95% CI 2-sided [-0.521 to 0.094]

30. Secondary Outcome: Change From Baseline in PGI-S Scores at Week 12
Description: as for outcome 27
Time Frame: Baseline, Week 12
Population: The ITT-RT comprised of all the subjects randomized at Visit 4.
Measure: Least Squares Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | FE 201836 500 ug (Randomized Treatment Period) | FE 201836 350 ug (Randomized Treatment Period) | FE 201836 250 ug (Randomized Treatment Period) | FE 201836 150 ug (Randomized Treatment Period) | FE 201836 100 ug (Randomized Treatment Period) | FE 201836 50 ug (Randomized Treatment Period) | Placebo (Randomized Treatment Period)
Number analyzed (Participants) | 45 | 22 | 18 | 13 | 12 | 27 | 70
score on a scale | -1.181 [-1.383 to -0.979] | -1.338 [-1.630 to -1.045] | -0.894 [-1.208 to -0.579] | -0.638 [-1.020 to -0.257] | -1.168 [-1.571 to -0.764] | -1.041 [-1.312 to -0.770] | -0.853 [-1.016 to -0.690]
Statistical Analysis 1: Comparison: FE 201836 500 ug (Randomized Treatment Period) vs Placebo (Randomized Treatment Period); Test type: Superiority; p = 0.0133, MMRM — Threshold for significance at 0.05 level; Least Square Mean Difference = -0.328, 95% CI 2-sided [-0.587 to -0.069]
Statistical Analysis 2: Comparison: FE 201836 350 ug (Randomized Treatment Period) vs Placebo (Randomized Treatment Period); Test type: Superiority; p = 0.0048, MMRM — Threshold for significance at 0.05 level; Least Square Mean Difference = -0.484, 95% CI 2-sided [-0.819 to -0.150]
Statistical Analysis 3: Comparison: FE 201836 250 ug (Randomized Treatment Period) vs Placebo (Randomized Treatment Period); Test type: Superiority; p = 0.8223, MMRM — Threshold for significance at 0.05 level; Least Square Mean Difference = -0.040, 95% CI 2-sided [-0.395 to 0.314]
Statistical Analysis 4: Comparison: FE 201836 150 ug (Randomized Treatment Period) vs Placebo (Randomized Treatment Period); Test type: Superiority; p = 0.3083, MMRM — Threshold for significance at 0.05 level; Least Square Mean Difference = 0.215, 95% CI 2-sided [-0.200 to 0.630]
Statistical Analysis 5: Comparison: FE 201836 100 ug (Randomized Treatment Period) vs Placebo (Randomized Treatment Period); Test type: Superiority; p = 0.1556, MMRM — Threshold for significance at 0.05 level; Least Square Mean Difference = -0.315, 95% CI 2-sided [-0.750 to 0.121]
Statistical Analysis 6: Comparison: FE 201836 50 ug (Randomized Treatment Period) vs Placebo (Randomized Treatment Period); Test type: Superiority; p = 0.2423, MMRM — Threshold for significance at 0.05 level; Least Square Mean Difference = -0.188, 95% CI 2-sided [-0.504 to 0.128]

31. Secondary Outcome: Change From Baseline in Hsu 5-point Likert Bother Scale at Week 1
Description: The Hsu 5-point Likert Bother scale is a questionnaire designed to assess the subjective bothersomeness and functional disruptiveness of nocturia. The Hsu 5 point Likert Bother Scale was scored from 0 (not at all) to 4 (extremely).
  Change from baseline in visit-specific Hsu Bother is presented in this endpoint.
  Level estimated for baseline value of Hsu Bother equal to 3 is presented in this endpoint.
Time Frame: Baseline, Week 1
Population: The ITT-RT comprised of all the subjects randomized at Visit 4.
Measure: Least Squares Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | FE 201836 500 ug (Randomized Treatment Period) | FE 201836 350 ug (Randomized Treatment Period) | FE 201836 250 ug (Randomized Treatment Period) | FE 201836 150 ug (Randomized Treatment Period) | FE 201836 100 ug (Randomized Treatment Period) | FE 201836 50 ug (Randomized Treatment Period) | Placebo (Randomized Treatment Period)
Number analyzed (Participants) | 50 | 23 | 24 | 14 | 9 | 30 | 70
score on a scale | -0.649 [-0.922 to -0.376] | -1.072 [-1.441 to -0.703] | -0.748 [-1.125 to -0.370] | -0.458 [-0.942 to 0.026] | -0.346 [-0.955 to 0.262] | -0.376 [-0.714 to -0.039] | -0.570 [-0.799 to -0.341]
Statistical Analysis 1: Comparison: FE 201836 500 ug (Randomized Treatment Period) vs Placebo (Randomized Treatment Period); Test type: Superiority; p = 0.6381, MMRM — Threshold for significance at 0.05 level; Least Square Mean Difference = -0.079, 95% CI 2-sided [-0.409 to 0.251]
Statistical Analysis 2: Comparison: FE 201836 350 ug (Randomized Treatment Period) vs Placebo (Randomized Treatment Period); Test type: Superiority; p = 0.0221, MMRM — Threshold for significance at 0.05 level; Least Square Mean Difference = -0.502, 95% CI 2-sided [-0.931 to -0.073]
Statistical Analysis 3: Comparison: FE 201836 250 ug (Randomized Treatment Period) vs Placebo (Randomized Treatment Period); Test type: Superiority; p = 0.4112, MMRM — Threshold for significance at 0.05 level; Least Square Mean Difference = -0.177, 95% CI 2-sided [-0.602 to 0.247]
Statistical Analysis 4: Comparison: FE 201836 150 ug (Randomized Treatment Period) vs Placebo (Randomized Treatment Period); Test type: Superiority; p = 0.6761, MMRM — Threshold for significance at 0.05 level; Least Square Mean Difference = 0.112, 95% CI 2-sided [-0.416 to 0.640]
Statistical Analysis 5: Comparison: FE 201836 100 ug (Randomized Treatment Period) vs Placebo (Randomized Treatment Period); Test type: Superiority; p = 0.4898, MMRM — Threshold for significance at 0.05 level; Least Square Mean Difference = 0.224, 95% CI 2-sided [-0.414 to 0.861]
Statistical Analysis 6: Comparison: FE 201836 50 ug (Randomized Treatment Period) vs Placebo (Randomized Treatment Period); Test type: Superiority; p = 0.3311, MMRM — Threshold for significance at 0.05 level; Least Square Mean Difference = 0.194, 95% CI 2-sided [-0.198 to 0.585]

32. Secondary Outcome: Change From Baseline in Hsu 5-point Likert Bother Scale at Week 4
Description: as for outcome 31
Time Frame: Baseline, Week 4
Population: The ITT-RT comprised of all the subjects randomized at Visit 4.
Measure: Least Squares Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | FE 201836 500 ug (Randomized Treatment Period) | FE 201836 350 ug (Randomized Treatment Period) | FE 201836 250 ug (Randomized Treatment Period) | FE 201836 150 ug (Randomized Treatment Period) | FE 201836 100 ug (Randomized Treatment Period) | FE 201836 50 ug (Randomized Treatment Period) | Placebo (Randomized Treatment Period)
Number analyzed (Participants) | 47 | 23 | 22 | 13 | 8 | 27 | 68
score on a scale | -0.896 [-1.161 to -0.630] | -0.940 [-1.294 to -0.586] | -0.712 [-1.083 to -0.340] | -0.606 [-1.079 to -0.132] | -1.096 [-1.698 to -0.493] | -0.861 [-1.193 to -0.530] | -0.665 [-0.885 to -0.445]
Statistical Analysis 1: Comparison: FE 201836 500 ug (Randomized Treatment Period) vs Placebo (Randomized Treatment Period); Test type: Superiority; p = 0.1583, MMRM — Threshold for significance at 0.05 level; Least Square Mean Difference = -0.230, 95% CI 2-sided [-0.551 to 0.090]
Statistical Analysis 2: Comparison: FE 201836 350 ug (Randomized Treatment Period) vs Placebo (Randomized Treatment Period); Test type: Superiority; p = 0.1884, MMRM — Threshold for significance at 0.05 level; Least Square Mean Difference = -0.275, 95% CI 2-sided [-0.685 to 0.136]
Statistical Analysis 3: Comparison: FE 201836 250 ug (Randomized Treatment Period) vs Placebo (Randomized Treatment Period); Test type: Superiority; p = 0.8256, MMRM — Threshold for significance at 0.05 level; Least Square Mean Difference = -0.047, 95% CI 2-sided [-0.463 to 0.369]
Statistical Analysis 4: Comparison: FE 201836 150 ug (Randomized Treatment Period) vs Placebo (Randomized Treatment Period); Test type: Superiority; p = 0.8198, MMRM — Threshold for significance at 0.05 level; Least Square Mean Difference = 0.059, 95% CI 2-sided [-0.455 to 0.574]
Statistical Analysis 5: Comparison: FE 201836 100 ug (Randomized Treatment Period) vs Placebo (Randomized Treatment Period); Test type: Superiority; p = 0.1793, MMRM — Threshold for significance at 0.05 level; Least Square Mean Difference = -0.431, 95% CI 2-sided [-1.061 to 0.199]
Statistical Analysis 6: Comparison: FE 201836 50 ug (Randomized Treatment Period) vs Placebo (Randomized Treatment Period); Test type: Superiority; p = 0.3155, MMRM — Threshold for significance at 0.05 level; Least Square Mean Difference = -0.196, 95% CI 2-sided [-0.581 to 0.189]

33. Secondary Outcome: Change From Baseline in Hsu 5-point Likert Bother Scale at Week 8
Description: as for outcome 31
Time Frame: Baseline, Week 8
Population: The ITT-RT comprised of all the subjects randomized at Visit 4.
Measure: Least Squares Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | FE 201836 500 ug (Randomized Treatment Period) | FE 201836 350 ug (Randomized Treatment Period) | FE 201836 250 ug (Randomized Treatment Period) | FE 201836 150 ug (Randomized Treatment Period) | FE 201836 100 ug (Randomized Treatment Period) | FE 201836 50 ug (Randomized Treatment Period) | Placebo (Randomized Treatment Period)
Number analyzed (Participants) | 40 | 24 | 23 | 14 | 7 | 27 | 71
score on a scale | -0.972 [-1.273 to -0.672] | -1.044 [-1.423 to -0.664] | -0.991 [-1.389 to -0.594] | -0.499 [-1.001 to 0.004] | -1.012 [-1.691 to -0.333] | -0.881 [-1.240 to -0.522] | -0.731 [-0.968 to -0.495]
Statistical Analysis 1: Comparison: FE 201836 500 ug (Randomized Treatment Period) vs Placebo (Randomized Treatment Period); Test type: Superiority; p = 0.1830, MMRM — Threshold for significance at 0.05 level; Least Square Mean Difference = -0.241, 95% CI 2-sided [-0.596 to 0.114]
Statistical Analysis 2: Comparison: FE 201836 350 ug (Randomized Treatment Period) vs Placebo (Randomized Treatment Period); Test type: Superiority; p = 0.1618, MMRM — Threshold for significance at 0.05 level; Least Square Mean Difference = -0.313, 95% CI 2-sided [-0.751 to 0.126]
Statistical Analysis 3: Comparison: FE 201836 250 ug (Randomized Treatment Period) vs Placebo (Randomized Treatment Period); Test type: Superiority; p = 0.2519, MMRM — Threshold for significance at 0.05 level; Least Square Mean Difference = -0.260, 95% CI 2-sided [-0.706 to 0.186]
Statistical Analysis 4: Comparison: FE 201836 150 ug (Randomized Treatment Period) vs Placebo (Randomized Treatment Period); Test type: Superiority; p = 0.4044, MMRM — Threshold for significance at 0.05 level; Least Square Mean Difference = 0.232, 95% CI 2-sided [-0.316 to 0.781]
Statistical Analysis 5: Comparison: FE 201836 100 ug (Randomized Treatment Period) vs Placebo (Randomized Treatment Period); Test type: Superiority; p = 0.4348, MMRM — Threshold for significance at 0.05 level; Least Square Mean Difference = -0.280, 95% CI 2-sided [-0.986 to 0.426]
Statistical Analysis 6: Comparison: FE 201836 50 ug (Randomized Treatment Period) vs Placebo (Randomized Treatment Period); Test type: Superiority; p = 0.4786, MMRM — Threshold for significance at 0.05 level; Least Square Mean Difference = -0.150, 95% CI 2-sided [-0.565 to 0.266]

34. Secondary Outcome: Change From Baseline in Hsu 5-point Likert Bother Scale at Week 12
Description: as for outcome 31
Time Frame: Baseline, Week 12
Population: The ITT-RT comprised of all the subjects randomized at Visit 4.
Measure: Least Squares Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | FE 201836 500 ug (Randomized Treatment Period) | FE 201836 350 ug (Randomized Treatment Period) | FE 201836 250 ug (Randomized Treatment Period) | FE 201836 150 ug (Randomized Treatment Period) | FE 201836 100 ug (Randomized Treatment Period) | FE 201836 50 ug (Randomized Treatment Period) | Placebo (Randomized Treatment Period)
Number analyzed (Participants) | 45 | 22 | 21 | 14 | 8 | 28 | 67
score on a scale | -0.992 [-1.306 to -0.679] | -1.249 [-1.663 to -0.834] | -0.700 [-1.132 to -0.267] | -0.880 [-1.416 to -0.343] | -0.974 [-1.676 to -0.272] | -0.921 [-1.303 to -0.540] | -0.769 [-1.027 to -0.511]
Statistical Analysis 1: Comparison: FE 201836 500 ug (Randomized Treatment Period) vs Placebo (Randomized Treatment Period); Test type: Superiority; p = 0.2412, MMRM — Threshold for significance at 0.05 level; Least Square Mean Difference = -0.223, 95% CI 2-sided [-0.598 to 0.151]
Statistical Analysis 2: Comparison: FE 201836 350 ug (Randomized Treatment Period) vs Placebo (Randomized Treatment Period); Test type: Superiority; p = 0.0501, MMRM — Threshold for significance at 0.05 level; Least Square Mean Difference = -0.480, 95% CI 2-sided [-0.959 to 0.000]
Statistical Analysis 3: Comparison: FE 201836 250 ug (Randomized Treatment Period) vs Placebo (Randomized Treatment Period); Test type: Superiority; p = 0.7788, MMRM — Threshold for significance at 0.05 level; Least Square Mean Difference = 0.069, 95% CI 2-sided [-0.417 to 0.556]
Statistical Analysis 4: Comparison: FE 201836 150 ug (Randomized Treatment Period) vs Placebo (Randomized Treatment Period); Test type: Superiority; p = 0.7111, MMRM — Threshold for significance at 0.05 level; Least Square Mean Difference = -0.111, 95% CI 2-sided [-0.698 to 0.477]
Statistical Analysis 5: Comparison: FE 201836 100 ug (Randomized Treatment Period) vs Placebo (Randomized Treatment Period); Test type: Superiority; p = 0.5816, MMRM — Threshold for significance at 0.05 level; Least Square Mean Difference = -0.205, 95% CI 2-sided [-0.937 to 0.527]
Statistical Analysis 6: Comparison: FE 201836 50 ug (Randomized Treatment Period) vs Placebo (Randomized Treatment Period); Test type: Superiority; p = 0.4981, MMRM — Threshold for significance at 0.05 level; Least Square Mean Difference = -0.152, 95% CI 2-sided [-0.595 to 0.290]

35. Secondary Outcome: Change From Baseline in ISI at Week 4
Description: The ISI is a 7-item questionnaire which comprises of four 'sleep-related' items and three 'wake-related' items. Each item is rated on a 0-4 scale and the total score ranges from 0 to 28 (higher score suggests more severe insomnia).
  Change from baseline in visit-specific ISI is presented in this endpoint.
  Level estimated for baseline value of ISI equal to 15 is presented in this endpoint.
Time Frame: Baseline, Week 4
Population: The ITT-RT comprised of all the subjects randomized at Visit 4.
Measure: Least Squares Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | FE 201836 500 ug (Randomized Treatment Period) | FE 201836 350 ug (Randomized Treatment Period) | FE 201836 250 ug (Randomized Treatment Period) | FE 201836 150 ug (Randomized Treatment Period) | FE 201836 100 ug (Randomized Treatment Period) | FE 201836 50 ug (Randomized Treatment Period) | Placebo (Randomized Treatment Period)
Number analyzed (Participants) | 47 | 24 | 22 | 13 | 8 | 27 | 68
score on a scale | -6.589 [-8.046 to -5.133] | -6.652 [-8.689 to -4.616] | -5.630 [-7.772 to -3.487] | -5.428 [-8.200 to -2.656] | -4.510 [-7.996 to -1.023] | -6.372 [-8.291 to -4.452] | -5.277 [-6.493 to -4.061]
Statistical Analysis 1: Comparison: FE 201836 500 ug (Randomized Treatment Period) vs Placebo (Randomized Treatment Period); Test type: Superiority; p = 0.1733, MMRM — Threshold for significance at 0.05 level; Least Square Mean Difference = -1.313, 95% CI 2-sided [-3.207 to 0.582]
Statistical Analysis 2: Comparison: FE 201836 350 ug (Randomized Treatment Period) vs Placebo (Randomized Treatment Period); Test type: Superiority; p = 0.2538, MMRM — Threshold for significance at 0.05 level; Least Square Mean Difference = -1.375, 95% CI 2-sided [-3.745 to 0.994]
Statistical Analysis 3: Comparison: FE 201836 250 ug (Randomized Treatment Period) vs Placebo (Randomized Treatment Period); Test type: Superiority; p = 0.7782, MMRM — Threshold for significance at 0.05 level; Least Square Mean Difference = -0.353, 95% CI 2-sided [-2.818 to 2.113]
Statistical Analysis 4: Comparison: FE 201836 150 ug (Randomized Treatment Period) vs Placebo (Randomized Treatment Period); Test type: Superiority; p = 0.9218, MMRM — Threshold for significance at 0.05 level; Least Square Mean Difference = -0.151, 95% CI 2-sided [-3.182 to 2.880]
Statistical Analysis 5: Comparison: FE 201836 100 ug (Randomized Treatment Period) vs Placebo (Randomized Treatment Period); Test type: Superiority; p = 0.6823, MMRM — Threshold for significance at 0.05 level; Least Square Mean Difference = 0.767, 95% CI 2-sided [-2.923 to 4.457]
Statistical Analysis 6: Comparison: FE 201836 50 ug (Randomized Treatment Period) vs Placebo (Randomized Treatment Period); Test type: Superiority; p = 0.3436, MMRM — Threshold for significance at 0.05 level; Least Square Mean Difference = -1.095, 95% CI 2-sided [-3.369 to 1.179]

36. Secondary Outcome: Change From Baseline in ISI at Week 8
Description: as for outcome 35
Time Frame: Baseline, Week 8
Population: The ITT-RT comprised of all the subjects randomized at Visit 4.
Measure: Least Squares Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | FE 201836 500 ug (Randomized Treatment Period) | FE 201836 350 ug (Randomized Treatment Period) | FE 201836 250 ug (Randomized Treatment Period) | FE 201836 150 ug (Randomized Treatment Period) | FE 201836 100 ug (Randomized Treatment Period) | FE 201836 50 ug (Randomized Treatment Period) | Placebo (Randomized Treatment Period)
Number analyzed (Participants) | 40 | 24 | 23 | 14 | 7 | 28 | 71
score on a scale | -7.643 [-9.140 to -6.147] | -8.091 [-10.116 to -6.067] | -6.693 [-8.799 to -4.588] | -6.959 [-9.668 to -4.250] | -5.707 [-9.283 to -2.131] | -7.167 [-9.055 to -5.280] | -6.408 [-7.603 to -5.213]
Statistical Analysis 1: Comparison: FE 201836 500 ug (Randomized Treatment Period) vs Placebo (Randomized Treatment Period); Test type: Superiority; p = 0.2042, MMRM — Threshold for significance at 0.05 level; Least Square Mean Difference = -1.235, 95% CI 2-sided [-3.146 to 0.676]
Statistical Analysis 2: Comparison: FE 201836 350 ug (Randomized Treatment Period) vs Placebo (Randomized Treatment Period); Test type: Superiority; p = 0.1591, MMRM — Threshold for significance at 0.05 level; Least Square Mean Difference = -1.683, 95% CI 2-sided [-4.031 to 0.665]
Statistical Analysis 3: Comparison: FE 201836 250 ug (Randomized Treatment Period) vs Placebo (Randomized Treatment Period); Test type: Superiority; p = 0.8168, MMRM — Threshold for significance at 0.05 level; Least Square Mean Difference = -0.285, 95% CI 2-sided [-2.708 to 2.138]
Statistical Analysis 4: Comparison: FE 201836 150 ug (Randomized Treatment Period) vs Placebo (Randomized Treatment Period); Test type: Superiority; p = 0.7148, MMRM — Threshold for significance at 0.05 level; Least Square Mean Difference = -0.551, 95% CI 2-sided [-3.517 to 2.416]
Statistical Analysis 5: Comparison: FE 201836 100 ug (Randomized Treatment Period) vs Placebo (Randomized Treatment Period); Test type: Superiority; p = 0.7141, MMRM — Threshold for significance at 0.05 level; Least Square Mean Difference = 0.701, 95% CI 2-sided [-3.066 to 4.468]
Statistical Analysis 6: Comparison: FE 201836 50 ug (Randomized Treatment Period) vs Placebo (Randomized Treatment Period); Test type: Superiority; p = 0.5041, MMRM — Threshold for significance at 0.05 level; Least Square Mean Difference = -0.759, 95% CI 2-sided [-2.995 to 1.477]

37. Secondary Outcome: Change From Baseline in ISI at Week 12
Description: as for outcome 35
Time Frame: Baseline, Week 12
Population: The ITT-RT comprised of all the subjects randomized at Visit 4.
Measure: Least Squares Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | FE 201836 500 ug (Randomized Treatment Period) | FE 201836 350 ug (Randomized Treatment Period) | FE 201836 250 ug (Randomized Treatment Period) | FE 201836 150 ug (Randomized Treatment Period) | FE 201836 100 ug (Randomized Treatment Period) | FE 201836 50 ug (Randomized Treatment Period) | Placebo (Randomized Treatment Period)
Number analyzed (Participants) | 45 | 22 | 21 | 14 | 8 | 27 | 67
score on a scale | -7.807 [-9.427 to -6.188] | -9.329 [-11.619 to -7.040] | -6.355 [-8.733 to -3.977] | -6.193 [-9.195 to -3.191] | -5.002 [-8.865 to -1.138] | -7.908 [-10.016 to -5.800] | -6.678 [-8.018 to -5.338]
Statistical Analysis 1: Comparison: FE 201836 500 ug (Randomized Treatment Period) vs Placebo (Randomized Treatment Period); Test type: Superiority; p = 0.2896, MMRM — Threshold for significance at 0.05 level; Least Square Mean Difference = -1.129, 95% CI 2-sided [-3.226 to 0.967]
Statistical Analysis 2: Comparison: FE 201836 350 ug (Randomized Treatment Period) vs Placebo (Randomized Treatment Period); Test type: Superiority; p = 0.0498, MMRM — Threshold for significance at 0.05 level; Least Square Mean Difference = -2.652, 95% CI 2-sided [-5.301 to -0.003]
Statistical Analysis 3: Comparison: FE 201836 250 ug (Randomized Treatment Period) vs Placebo (Randomized Treatment Period); Test type: Superiority; p = 0.8159, MMRM — Threshold for significance at 0.05 level; Least Square Mean Difference = 0.323, 95% CI 2-sided [-2.409 to 3.055]
Statistical Analysis 4: Comparison: FE 201836 150 ug (Randomized Treatment Period) vs Placebo (Randomized Treatment Period); Test type: Superiority; p = 0.7719, MMRM — Threshold for significance at 0.05 level; Least Square Mean Difference = 0.485, 95% CI 2-sided [-2.809 to 3.779]
Statistical Analysis 5: Comparison: FE 201836 100 ug (Randomized Treatment Period) vs Placebo (Randomized Treatment Period); Test type: Superiority; p = 0.4193, MMRM — Threshold for significance at 0.05 level; Least Square Mean Difference = 1.676, 95% CI 2-sided [-2.407 to 5.760]
Statistical Analysis 6: Comparison: FE 201836 50 ug (Randomized Treatment Period) vs Placebo (Randomized Treatment Period); Test type: Superiority; p = 0.3333, MMRM — Threshold for significance at 0.05 level; Least Square Mean Difference = -1.230, 95% CI 2-sided [-3.730 to 1.270]

38. Secondary Outcome: Change From Baseline in Mean Duration of First Undisturbed Sleep Period (FUSP) at Week 1
Description: The FUSP is defined as the time in minutes from the time of going to bed to the time of first nocturnal void, or time of awakening if no void occured.
  The duration of FUSP at each visit was calculated as the average over the 3 consecutive 24-hour periods just prior to the respective visit. Adjusted visit-specific mean changes from baseline in FUSP are estimated using a baseline value of 180 (min).
Time Frame: Baseline, Week 1
Population: The ITT-RT comprised of all the subjects randomized at Visit 4.
Measure: Mean (95% Confidence Interval); unit: minutes
Arm/Group | FE 201836 500 ug (Randomized Treatment Period) | FE 201836 350 ug (Randomized Treatment Period) | FE 201836 250 ug (Randomized Treatment Period) | FE 201836 150 ug (Randomized Treatment Period) | FE 201836 100 ug (Randomized Treatment Period) | FE 201836 50 ug (Randomized Treatment Period) | Placebo (Randomized Treatment Period)
Number analyzed (Participants) | 54 | 24 | 24 | 14 | 11 | 33 | 80
minutes | 122.9 [86.2 to 159.7] | 187.0 [132.3 to 241.7] | 106.0 [49.6 to 162.4] | 91.7 [18.7 to 164.8] | 82.9 [2.5 to 163.4] | 51.3 [3.9 to 98.7] | 81.1 [50.8 to 111.4]
Statistical Analysis 1: Comparison: FE 201836 500 ug (Randomized Treatment Period) vs Placebo (Randomized Treatment Period); Test type: Superiority; p = 0.0853, MMRM — Threshold for significance at 0.05 level; Mean Difference = 41.8, 95% CI 2-sided [-5.9 to 89.6]
Statistical Analysis 2: Comparison: FE 201836 350 ug (Randomized Treatment Period) vs Placebo (Randomized Treatment Period); Test type: Superiority; p = 0.0010, MMRM — Threshold for significance at 0.05 level; Mean Difference = 105.9, 95% CI 2-sided [43.4 to 168.4]
Statistical Analysis 3: Comparison: FE 201836 250 ug (Randomized Treatment Period) vs Placebo (Randomized Treatment Period); Test type: Superiority; p = 0.4418, MMRM — Threshold for significance at 0.05 level; Mean Difference = 24.9, 95% CI 2-sided [-38.8 to 88.6]
Statistical Analysis 4: Comparison: FE 201836 150 ug (Randomized Treatment Period) vs Placebo (Randomized Treatment Period); Test type: Superiority; p = 0.7902, MMRM — Threshold for significance at 0.05 level; Mean Difference = 10.7, 95% CI 2-sided [-68.2 to 89.6]
Statistical Analysis 5: Comparison: FE 201836 100 ug (Randomized Treatment Period) vs Placebo (Randomized Treatment Period); Test type: Superiority; p = 0.9664, MMRM — Threshold for significance at 0.05 level; Mean Difference = 1.8, 95% CI 2-sided [-84.2 to 87.9]
Statistical Analysis 6: Comparison: FE 201836 50 ug (Randomized Treatment Period) vs Placebo (Randomized Treatment Period); Test type: Superiority; p = 0.2977, MMRM — Threshold for significance at 0.05 level; Mean Difference = -29.8, 95% CI 2-sided [-85.9 to 26.4]

39. Secondary Outcome: Change From Baseline in Mean Duration of FUSP at Week 4
Description: The FUSP is defined as the time in minutes from the time of going to bed to the time of first nocturnal void, or time of awakening if no void occurred.
  The duration of FUSP at each visit was calculated as the average over the 3 consecutive 24-hour periods just prior to the respective visit. Adjusted visit-specific mean changes from baseline in FUSP are estimated using a baseline value of 180 (min).
Time Frame: Baseline, Week 4
Population: The ITT-RT comprised of all the subjects randomized at Visit 4.
Measure: Mean (95% Confidence Interval); unit: minutes
Arm/Group | FE 201836 500 ug (Randomized Treatment Period) | FE 201836 350 ug (Randomized Treatment Period) | FE 201836 250 ug (Randomized Treatment Period) | FE 201836 150 ug (Randomized Treatment Period) | FE 201836 100 ug (Randomized Treatment Period) | FE 201836 50 ug (Randomized Treatment Period) | Placebo (Randomized Treatment Period)
Number analyzed (Participants) | 50 | 22 | 21 | 12 | 12 | 31 | 76
minutes | 164.5 [127.9 to 201.0] | 211.0 [156.3 to 265.7] | 132.3 [75.2 to 189.4] | 89.5 [15.1 to 163.9] | 122.0 [46.8 to 197.3] | 95.5 [48.6 to 142.5] | 150.2 [120.4 to 180.0]
Statistical Analysis 1: Comparison: FE 201836 500 ug (Randomized Treatment Period) vs Placebo (Randomized Treatment Period); Test type: Superiority; p = 0.5523, MMRM — Threshold for significance at 0.05 level; Mean Difference = 14.3, 95% CI 2-sided [-33.0 to 61.5]
Statistical Analysis 2: Comparison: FE 201836 350 ug (Randomized Treatment Period) vs Placebo (Randomized Treatment Period); Test type: Superiority; p = 0.0556, MMRM — Threshold for significance at 0.05 level; Mean Difference = 60.8, 95% CI 2-sided [-1.5 to 123.0]
Statistical Analysis 3: Comparison: FE 201836 250 ug (Randomized Treatment Period) vs Placebo (Randomized Treatment Period); Test type: Superiority; p = 0.5837, MMRM — Threshold for significance at 0.05 level; Mean Difference = -17.9, 95% CI 2-sided [-82.0 to 46.3]
Statistical Analysis 4: Comparison: FE 201836 150 ug (Randomized Treatment Period) vs Placebo (Randomized Treatment Period); Test type: Superiority; p = 0.1363, MMRM — Threshold for significance at 0.05 level; Mean Difference = -60.7, 95% CI 2-sided [-140.7 to 19.3]
Statistical Analysis 5: Comparison: FE 201836 100 ug (Randomized Treatment Period) vs Placebo (Randomized Treatment Period); Test type: Superiority; p = 0.4938, MMRM — Threshold for significance at 0.05 level; Mean Difference = -28.2, 95% CI 2-sided [-109.1 to 52.8]
Statistical Analysis 6: Comparison: FE 201836 50 ug (Randomized Treatment Period) vs Placebo (Randomized Treatment Period); Test type: Superiority; p = 0.0535, MMRM — Threshold for significance at 0.05 level; Mean Difference = -54.7, 95% CI 2-sided [-110.2 to 0.8]

40. Secondary Outcome: Change From Baseline in Mean Duration of FUSP at Week 8
Description: as for outcome 39
Time Frame: Baseline, Week 8
Population: The ITT-RT comprised of all the subjects randomized at Visit 4.
Measure: Mean (95% Confidence Interval); unit: minutes
Arm/Group | FE 201836 500 ug (Randomized Treatment Period) | FE 201836 350 ug (Randomized Treatment Period) | FE 201836 250 ug (Randomized Treatment Period) | FE 201836 150 ug (Randomized Treatment Period) | FE 201836 100 ug (Randomized Treatment Period) | FE 201836 50 ug (Randomized Treatment Period) | Placebo (Randomized Treatment Period)
Number analyzed (Participants) | 44 | 23 | 21 | 14 | 12 | 30 | 70
minutes | 160.4 [112.4 to 208.3] | 225.4 [157.9 to 293.0] | 190.2 [118.9 to 261.6] | 136.8 [48.3 to 225.4] | 163.2 [68.7 to 257.8] | 164.3 [104.9 to 223.7] | 161.0 [122.6 to 199.5]
Statistical Analysis 1: Comparison: FE 201836 500 ug (Randomized Treatment Period) vs Placebo (Randomized Treatment Period); Test type: Superiority; p = 0.9829, MMRM — Threshold for significance at 0.05 level; Mean Difference = -0.7, 95% CI 2-sided [-62.2 to 60.9]
Statistical Analysis 2: Comparison: FE 201836 350 ug (Randomized Treatment Period) vs Placebo (Randomized Treatment Period); Test type: Superiority; p = 0.1038, MMRM — Threshold for significance at 0.05 level; Mean Difference = 64.4, 95% CI 2-sided [-13.3 to 142.1]
Statistical Analysis 3: Comparison: FE 201836 250 ug (Randomized Treatment Period) vs Placebo (Randomized Treatment Period); Test type: Superiority; p = 0.4764, MMRM — Threshold for significance at 0.05 level; Mean Difference = 29.2, 95% CI 2-sided [-51.4 to 109.8]
Statistical Analysis 4: Comparison: FE 201836 150 ug (Randomized Treatment Period) vs Placebo (Randomized Treatment Period); Test type: Superiority; p = 0.6204, MMRM — Threshold for significance at 0.05 level; Mean Difference = -24.2, 95% CI 2-sided [-120.5 to 72.0]
Statistical Analysis 5: Comparison: FE 201836 100 ug (Randomized Treatment Period) vs Placebo (Randomized Treatment Period); Test type: Superiority; p = 0.9660, MMRM — Threshold for significance at 0.05 level; Mean Difference = 2.2, 95% CI 2-sided [-100.1 to 104.6]
Statistical Analysis 6: Comparison: FE 201836 50 ug (Randomized Treatment Period) vs Placebo (Randomized Treatment Period); Test type: Superiority; p = 0.9275, MMRM — Threshold for significance at 0.05 level; Mean Difference = 3.3, 95% CI 2-sided [-67.4 to 73.9]

41. Secondary Outcome: Change From Baseline in Mean Duration of FUSP at Week 12
Description: as for outcome 39
Time Frame: Baseline, Week 12
Population: The ITT-RT comprised of all the subjects randomized at Visit 4.
Measure: Mean (95% Confidence Interval); unit: minutes
Arm/Group | FE 201836 500 ug (Randomized Treatment Period) | FE 201836 350 ug (Randomized Treatment Period) | FE 201836 250 ug (Randomized Treatment Period) | FE 201836 150 ug (Randomized Treatment Period) | FE 201836 100 ug (Randomized Treatment Period) | FE 201836 50 ug (Randomized Treatment Period) | Placebo (Randomized Treatment Period)
Number analyzed (Participants) | 40 | 19 | 19 | 14 | 11 | 29 | 69
minutes | 178.5 [132.5 to 224.5] | 160.0 [93.3 to 226.6] | 180.7 [112.2 to 249.2] | 111.5 [29.7 to 193.2] | 141.1 [51.3 to 230.9] | 166.2 [110.5 to 221.8] | 162.8 [126.9 to 198.7]
Statistical Analysis 1: Comparison: FE 201836 500 ug (Randomized Treatment Period) vs Placebo (Randomized Treatment Period); Test type: Superiority; p = 0.5964, MMRM — Threshold for significance at 0.05 level; Mean Difference = 15.7, 95% CI 2-sided [-42.7 to 74.2]
Statistical Analysis 2: Comparison: FE 201836 350 ug (Randomized Treatment Period) vs Placebo (Randomized Treatment Period); Test type: Superiority; p = 0.9418, MMRM — Threshold for significance at 0.05 level; Mean Difference = -2.8, 95% CI 2-sided [-78.5 to 72.9]
Statistical Analysis 3: Comparison: FE 201836 250 ug (Randomized Treatment Period) vs Placebo (Randomized Treatment Period); Test type: Superiority; p = 0.6452, MMRM — Threshold for significance at 0.05 level; Mean Difference = 18.0, 95% CI 2-sided [-58.8 to 94.7]
Statistical Analysis 4: Comparison: FE 201836 150 ug (Randomized Treatment Period) vs Placebo (Randomized Treatment Period); Test type: Superiority; p = 0.2565, MMRM — Threshold for significance at 0.05 level; Mean Difference = -51.3, 95% CI 2-sided [-140.2 to 37.6]
Statistical Analysis 5: Comparison: FE 201836 100 ug (Randomized Treatment Period) vs Placebo (Randomized Treatment Period); Test type: Other; p = 0.6605, MMRM — Threshold for significance at 0.05 level; Mean Difference = -21.6, 95% CI 2-sided [-118.6 to 75.4]
Statistical Analysis 6: Comparison: FE 201836 50 ug (Randomized Treatment Period) vs Placebo (Randomized Treatment Period); Test type: Superiority; p = 0.9191, MMRM — Threshold for significance at 0.05 level; Mean Difference = 3.4, 95% CI 2-sided [-62.6 to 69.4]

42. Secondary Outcome: Change From Baseline in Aggregated Mean Duration of FUSP During 12 Weeks of Treatment
Description: The FUSP is defined as the time in minutes from the time of going to bed to the time of first nocturnal void, or time of awakening if no void occurred.
  The visit-specific means were aggregated into a mean of current and preceding visits.
  Level estimated for baseline value of mean duration of FUSP (minutes) equal to 180 is presented in this endpoint.
  The 95% credibility interval (2.5 and 97.5 percentiles of the posterior distribution) instead of confidence interval is presented for this endpoint.
Time Frame: Baseline, During 12 Weeks of Treatment
Population: The ITT-RT comprised of all the subjects randomized at Visit 4.
Measure: Mean (95% Confidence Interval); unit: minutes
Arm/Group | FE 201836 500 ug (Randomized Treatment Period) | FE 201836 350 ug (Randomized Treatment Period) | FE 201836 250 ug (Randomized Treatment Period) | FE 201836 150 ug (Randomized Treatment Period) | FE 201836 100 ug (Randomized Treatment Period) | FE 201836 50 ug (Randomized Treatment Period) | Placebo (Randomized Treatment Period)
Number analyzed (Participants) | 60 | 27 | 24 | 14 | 13 | 34 | 87
minutes | 154.98 [130.41 to 189.10] | 150.23 [130.20 to 181.15] | 145.95 [128.21 to 170.90] | 140.74 [120.51 to 160.16] | 139.19 [117.86 to 157.42] | 138.13 [115.62 to 157.24] | 137.45 [114.12 to 157.30]
Statistical Analysis 1: Comparison: FE 201836 500 ug (Randomized Treatment Period) vs Placebo (Randomized Treatment Period); Based on a Bayesian analysis of a sigmoidal dose-response relationship; Test type: Superiority; Mean Difference = 17.52, 95% CI 2-sided [-6.19 to 62.09]
Statistical Analysis 2: Comparison: FE 201836 350 ug (Randomized Treatment Period) vs Placebo (Randomized Treatment Period); Based on a Bayesian analysis of a sigmoidal dose-response relationship; Test type: Superiority; Mean Difference = 12.78, 95% CI 2-sided [-0.73 to 55.89]
Statistical Analysis 3: Comparison: FE 201836 250 ug (Randomized Treatment Period) vs Placebo (Randomized Treatment Period); Based on a Bayesian analysis of a sigmoidal dose-response relationship; Test type: Superiority; Mean Difference = 8.50, 95% CI 2-sided [-0.14 to 47.28]
Statistical Analysis 4: Comparison: FE 201836 150 ug (Randomized Treatment Period) vs Placebo (Randomized Treatment Period); Based on a Bayesian analysis of a sigmoidal dose-response relationship; Test type: Superiority; Mean Difference = 3.29, 95% CI 2-sided [-0.01 to 28.07]
Statistical Analysis 5: Comparison: FE 201836 100 ug (Randomized Treatment Period) vs Placebo (Randomized Treatment Period); Based on a Bayesian analysis of a sigmoidal dose-response relationship; Test type: Superiority; Mean Difference = 1.74, 95% CI 2-sided [-0.00 to 17.90]
Statistical Analysis 6: Comparison: FE 201836 50 ug (Randomized Treatment Period) vs Placebo (Randomized Treatment Period); Based on a Bayesian analysis of a sigmoidal dose-response relationship; Test type: Superiority; Mean Difference = 0.68, 95% CI 2-sided [-0.00 to 7.55]

43. Secondary Outcome: Change From Baseline in Nocturnal Diuresis Rate Profiles at Week 1
Description: The nocturnal diuresis rate (mL/min) is calculated as the mean of the nocturnal diuresis for each of the three nights, with the single-night nocturnal diuresis calculated as the ratio of NUV to total time in bed.
  Change from baseline in visit-specific mean nocturnal diuresis (mL/min) is presented.
  Level estimated for baseline value of mean nocturnal diuresis (mL/min) equal to 1.3 is presented in this endpoint.
Time Frame: Baseline, Week 1
Population: The ITT-RT comprised of all the subjects randomized at Visit 4.
Measure: Mean (95% Confidence Interval); unit: mL/min
Arm/Group | FE 201836 500 ug (Randomized Treatment Period) | FE 201836 350 ug (Randomized Treatment Period) | FE 201836 250 ug (Randomized Treatment Period) | FE 201836 150 ug (Randomized Treatment Period) | FE 201836 100 ug (Randomized Treatment Period) | FE 201836 50 ug (Randomized Treatment Period) | Placebo (Randomized Treatment Period)
Number analyzed (Participants) | 53 | 24 | 24 | 14 | 11 | 32 | 78
mL/min | -0.575 [-0.687 to -0.463] | -0.635 [-0.801 to -0.468] | -0.610 [-0.779 to -0.440] | -0.459 [-0.678 to -0.239] | -0.523 [-0.766 to -0.280] | -0.328 [-0.474 to -0.182] | -0.402 [-0.494 to -0.310]
Statistical Analysis 1: Comparison: FE 201836 500 ug (Randomized Treatment Period) vs Placebo (Randomized Treatment Period); Test type: Superiority; p = 0.0196, MMRM — Threshold for significance at 0.05 level; Mean Difference = -0.173, 95% CI 2-sided [-0.318 to -0.028]
Statistical Analysis 2: Comparison: FE 201836 350 ug (Randomized Treatment Period) vs Placebo (Randomized Treatment Period); Test type: Superiority; p = 0.0167, MMRM — Threshold for significance at 0.05 level; Mean Difference = -0.233, 95% CI 2-sided [-0.423 to -0.043]
Statistical Analysis 3: Comparison: FE 201836 250 ug (Randomized Treatment Period) vs Placebo (Randomized Treatment Period); Test type: Superiority; p = 0.0352, MMRM — Threshold for significance at 0.05 level; Mean Difference = -0.208, 95% CI 2-sided [-0.401 to -0.015]
Statistical Analysis 4: Comparison: FE 201836 150 ug (Randomized Treatment Period) vs Placebo (Randomized Treatment Period); Test type: Superiority; p = 0.6402, MMRM — Threshold for significance at 0.05 level; Mean Difference = -0.057, 95% CI 2-sided [-0.295 to 0.182]
Statistical Analysis 5: Comparison: FE 201836 100 ug (Randomized Treatment Period) vs Placebo (Randomized Treatment Period); Test type: Superiority; p = 0.3602, MMRM — Threshold for significance at 0.05 level; Mean Difference = -0.121, 95% CI 2-sided [-0.381 to 0.139]
Statistical Analysis 6: Comparison: FE 201836 50 ug (Randomized Treatment Period) vs Placebo (Randomized Treatment Period); Test type: Superiority; p = 0.4018, MMRM — Threshold for significance at 0.05 level; Mean Difference = 0.074, 95% CI 2-sided [-0.099 to 0.247]

44. Secondary Outcome: Change From Baseline in Nocturnal Diuresis Rate Profiles at Week 12
Description: as for outcome 43
Time Frame: Baseline, Week 12
Population: The ITT-RT comprised of all the subjects randomized at Visit 4.
Measure: Mean (95% Confidence Interval); unit: mL/min
Arm/Group | FE 201836 500 ug (Randomized Treatment Period) | FE 201836 350 ug (Randomized Treatment Period) | FE 201836 250 ug (Randomized Treatment Period) | FE 201836 150 ug (Randomized Treatment Period) | FE 201836 100 ug (Randomized Treatment Period) | FE 201836 50 ug (Randomized Treatment Period) | Placebo (Randomized Treatment Period)
Number analyzed (Participants) | 35 | 18 | 18 | 14 | 11 | 29 | 68
mL/min | -0.648 [-0.789 to -0.508] | -0.606 [-0.805 to -0.408] | -0.735 [-0.937 to -0.533] | -0.458 [-0.693 to -0.223] | -0.685 [-0.945 to -0.425] | -0.651 [-0.812 to -0.490] | -0.515 [-0.619 to -0.412]
Statistical Analysis 1: Comparison: FE 201836 500 ug (Randomized Treatment Period) vs Placebo (Randomized Treatment Period); Test type: Superiority; p = 0.1354, MMRM — Threshold for significance at 0.05 level; Mean Difference = -0.133, 95% CI 2-sided [-0.308 to 0.042]
Statistical Analysis 2: Comparison: FE 201836 350 ug (Randomized Treatment Period) vs Placebo (Randomized Treatment Period); Test type: Superiority; p = 0.4238, MMRM — Threshold for significance at 0.05 level; Mean Difference = -0.091, 95% CI 2-sided [-0.315 to 0.133]
Statistical Analysis 3: Comparison: FE 201836 250 ug (Randomized Treatment Period) vs Placebo (Randomized Treatment Period); Test type: Superiority; p = 0.0574, MMRM — Threshold for significance at 0.05 level; Mean Difference = -0.220, 95% CI 2-sided [-0.446 to 0.007]
Statistical Analysis 4: Comparison: FE 201836 150 ug (Randomized Treatment Period) vs Placebo (Randomized Treatment Period); Test type: Superiority; p = 0.6579, MMRM — Threshold for significance at 0.05 level; Mean Difference = 0.058, 95% CI 2-sided [-0.199 to 0.315]
Statistical Analysis 5: Comparison: FE 201836 100 ug (Randomized Treatment Period) vs Placebo (Randomized Treatment Period); Test type: Superiority; p = 0.2337, MMRM — Threshold for significance at 0.05 level; Mean Difference = -0.170, 95% CI 2-sided [-0.450 to 0.110]
Statistical Analysis 6: Comparison: FE 201836 50 ug (Randomized Treatment Period) vs Placebo (Randomized Treatment Period); Test type: Superiority; p = 0.1639, MMRM — Threshold for significance at 0.05 level; Mean Difference = -0.136, 95% CI 2-sided [-0.328 to 0.056]

45. Secondary Outcome: Change From Baseline in Mean NUV in Week 1
Description: The NUV is defined as the total urine volume from 5 minutes after bedtime with the intention to sleep including the first void within 30 minutes of rising in the morning.
  The NUV at each visit was calculated as the average over the 3 consecutive 24-hour periods just prior to the respective visit. Adjusted visit-specific mean changes from baseline in NUV are estimated using a baseline value of 750 (mL).
Time Frame: Baseline, Week 1
Population: The ITT-RT comprised of all the subjects randomized at Visit 4.
Measure: Mean (95% Confidence Interval); unit: mL
Arm/Group | FE 201836 500 ug (Randomized Treatment Period) | FE 201836 350 ug (Randomized Treatment Period) | FE 201836 250 ug (Randomized Treatment Period) | FE 201836 150 ug (Randomized Treatment Period) | FE 201836 100 ug (Randomized Treatment Period) | FE 201836 50 ug (Randomized Treatment Period) | Placebo (Randomized Treatment Period)
Number analyzed (Participants) | 53 | 24 | 24 | 14 | 11 | 32 | 78
mL | -328.8 [-395.3 to -262.3] | -371.8 [-470.4 to -273.3] | -352.4 [-452.8 to -252.1] | -265.5 [-395.5 to -135.6] | -312.6 [-455.9 to -169.3] | -218.2 [-304.9 to -131.6] | -241.6 [-296.3 to -186.9]
Statistical Analysis 1: Comparison: FE 201836 500 ug (Randomized Treatment Period) vs Placebo (Randomized Treatment Period); Test type: Superiority; p = 0.0470, MMRM; Mean Difference = -87.2, 95% CI 2-sided [-173.2 to -1.2]
Statistical Analysis 2: Comparison: FE 201836 350 ug (Randomized Treatment Period) vs Placebo (Randomized Treatment Period); Test type: Superiority; p = 0.0237, MMRM; Mean Difference = -130.2, 95% CI 2-sided [-242.9 to -17.6]
Statistical Analysis 3: Comparison: FE 201836 250 ug (Randomized Treatment Period) vs Placebo (Randomized Treatment Period); Test type: Superiority; p = 0.0569, MMRM; Mean Difference = -110.8, 95% CI 2-sided [-224.9 to 3.3]
Statistical Analysis 4: Comparison: FE 201836 150 ug (Randomized Treatment Period) vs Placebo (Randomized Treatment Period); Test type: Superiority; p = 0.7383, MMRM; Mean Difference = -23.9, 95% CI 2-sided [-164.8 to 117.0]
Statistical Analysis 5: Comparison: FE 201836 100 ug (Randomized Treatment Period) vs Placebo (Randomized Treatment Period); Test type: Superiority; p = 0.3626, MMRM; Mean Difference = -71.0, 95% CI 2-sided [-224.3 to 82.3]
Statistical Analysis 6: Comparison: FE 201836 50 ug (Randomized Treatment Period) vs Placebo (Randomized Treatment Period); Test type: Superiority; p = 0.6524, MMRM; Mean Difference = 23.4, 95% CI 2-sided [-78.9 to 125.7]

46. Secondary Outcome: Change From Baseline in Mean NUV at Week 12
Description: as for outcome 45
Time Frame: Baseline, Week 12
Population: The ITT-RT comprised of all the subjects randomized at Visit 4.
Measure: Mean (95% Confidence Interval); unit: mL
Arm/Group | FE 201836 500 ug (Randomized Treatment Period) | FE 201836 350 ug (Randomized Treatment Period) | FE 201836 250 ug (Randomized Treatment Period) | FE 201836 150 ug (Randomized Treatment Period) | FE 201836 100 ug (Randomized Treatment Period) | FE 201836 50 ug (Randomized Treatment Period) | Placebo (Randomized Treatment Period)
Number analyzed (Participants) | 35 | 18 | 18 | 14 | 11 | 29 | 68
mL | -367.3 [-447.1 to -287.5] | -392.4 [-505.2 to -279.5] | -411.3 [-526.0 to -296.7] | -284.2 [-418.4 to -149.9] | -393.5 [-541.9 to -245.1] | -403.2 [-495.5 to -310.9] | -317.8 [-377.1 to -258.5]
Statistical Analysis 1: Comparison: FE 201836 500 ug (Randomized Treatment Period) vs Placebo (Randomized Treatment Period); Test type: Superiority; p = 0.3273, MMRM — Threshold for significance at 0.05 level; Mean Difference = -49.5, 95% CI 2-sided [-148.9 to 49.9]
Statistical Analysis 2: Comparison: FE 201836 350 ug (Randomized Treatment Period) vs Placebo (Randomized Treatment Period); Test type: Superiority; p = 0.2500, MMRM — Threshold for significance at 0.05 level; Mean Difference = -74.6, 95% CI 2-sided [-202.0 to 52.9]
Statistical Analysis 3: Comparison: FE 201836 250 ug (Randomized Treatment Period) vs Placebo (Randomized Treatment Period); Test type: Superiority; p = 0.1537, MMRM — Threshold for significance at 0.05 level; Mean Difference = -93.5, 95% CI 2-sided [-222.3 to 35.2]
Statistical Analysis 4: Comparison: FE 201836 150 ug (Randomized Treatment Period) vs Placebo (Randomized Treatment Period); Test type: Superiority; p = 0.6515, MMRM — Threshold for significance at 0.05 level; Mean Difference = 33.6, 95% CI 2-sided [-113.1 to 180.3]
Statistical Analysis 5: Comparison: FE 201836 100 ug (Randomized Treatment Period) vs Placebo (Randomized Treatment Period); Test type: Superiority; p = 0.3506, MMRM — Threshold for significance at 0.05 level; Mean Difference = -75.7, 95% CI 2-sided [-235.3 to 83.9]
Statistical Analysis 6: Comparison: FE 201836 50 ug (Randomized Treatment Period) vs Placebo (Randomized Treatment Period); Test type: Superiority; p = 0.1255, MMRM — Threshold for significance at 0.05 level; Mean Difference = -85.4, 95% CI 2-sided [-194.8 to 24.1]

ADVERSE EVENTS:
Time Frame: Enrichment period: Treatment-emergent adverse events (AEs) occurring in the time interval from V2 (active run-in) to V4 (randomization), including AEs with missing start date. Randomized treatment period: Treatment-emergent AEs occurring in the time interval from V4 to end-of-trial.
Description: The Safety Analysis Set for the enrichment period comprised subjects who received investigational medicinal product (IMP) at V2 and did not return all IMP unused at/before V4. The Safety Analysis Set for the randomized treatment period comprised subjects who received IMP at V4 and did not return all IMP unused, and who had at least 1 safety assessment after V4.
Groups:
- FE 201836 500 µg (Enrichment Period); FE 201836 500 µg (Randomized Treatment Period): FE 201836 500 µg oral solution and placebo ODT, administered once daily
Arm/Group | FE 201836 500 µg (Enrichment Period) | FE 201836 500 µg (Randomized Treatment Period) | FE 201836 350 µg (Randomized Treatment Period) | FE 201836 250 µg (Randomized Treatment Period) | FE 201836 150 µg (Randomized Treatment Period) | FE 201836 100 µg (Randomized Treatment Period) | FE 201836 50 µg (Randomized Treatment Period) | Placebo (Randomized Treatment Period) | Desmopressin 25 µg (Randomized Treatment Period) | Desmopressin 50 µg (Randomized Treatment Period)
All-Cause Mortality (participants affected / at risk) | 0/531 | 0/60 | 0/27 | 0/24 | 0/14 | 0/13 | 0/34 | 0/87 | 0/26 | 0/17
Serious Adverse Events (participants affected / at risk) | 2/531 | 1/60 | 2/27 | 1/24 | 0/14 | 1/13 | 0/34 | 2/87 | 0/26 | 0/17
Other Adverse Events (participants affected / at risk) | 0/531 | 16/60 | 3/27 | 3/24 | 8/14 | 5/13 | 7/34 | 16/87 | 8/26 | 9/17
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | FE 201836 500 µg (Enrichment Period) (N=531) | FE 201836 500 µg (Randomized Treatment Period) (N=60) | FE 201836 350 µg (Randomized Treatment Period) (N=27) | FE 201836 250 µg (Randomized Treatment Period) (N=24) | FE 201836 150 µg (Randomized Treatment Period) (N=14) | FE 201836 100 µg (Randomized Treatment Period) (N=13) | FE 201836 50 µg (Randomized Treatment Period) (N=34) | Placebo (Randomized Treatment Period) (N=87) | Desmopressin 25 µg (Randomized Treatment Period) (N=26) | Desmopressin 50 µg (Randomized Treatment Period) (N=17)
Hyponatraemia (Metabolism and nutrition disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Colitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Serum sickness-like reaction (Immune system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastroenteritis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Staphylococcal infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Transitional cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Syncope (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Urticaria (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Facial bones fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Subdural haematoma (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | FE 201836 500 µg (Enrichment Period) (N=531) | FE 201836 500 µg (Randomized Treatment Period) (N=60) | FE 201836 350 µg (Randomized Treatment Period) (N=27) | FE 201836 250 µg (Randomized Treatment Period) (N=24) | FE 201836 150 µg (Randomized Treatment Period) (N=14) | FE 201836 100 µg (Randomized Treatment Period) (N=13) | FE 201836 50 µg (Randomized Treatment Period) (N=34) | Placebo (Randomized Treatment Period) (N=87) | Desmopressin 25 µg (Randomized Treatment Period) (N=26) | Desmopressin 50 µg (Randomized Treatment Period) (N=17)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Vertigo (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (3)
Nausea (Gastrointestinal disorders) | 0 (0) | 3 (3) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 3 (4) | 0 (0) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Urinary tract infection (Infections and infestations) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cellulitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Accidental overdose (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 3 (4) | 0 (0) | 4 (6)
Hand fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Laceration (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Road traffic accident (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Weight increased (Investigations) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Gamma-glutamyltransferase increased (Investigations) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood creatine phosphokinase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Blood sodium decreased (Investigations) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Hepatic enzyme increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0)
Alanine aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood alkaline phosphatase (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 0 (0) | 3 (5) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypoglycaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Joint swelling (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 0 (0) | 3 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 1 (1) | 0 (0)
Insomnia (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Dysuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Renal impairment (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (2) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other

DOCUMENTS (2):
  • Study Protocol (2018-07-05): https://cdn.clinicaltrials.gov/large-docs/19/NCT03201419/Prot_000.pdf
  • Statistical Analysis Plan (2019-12-12): https://cdn.clinicaltrials.gov/large-docs/19/NCT03201419/SAP_001.pdf